CLINICAL TRIAL: NCT03235726
Title: A Double-blind (Sponsor Unblind), Randomized, Placebo-controlled, Single and Repeat Escalating Dose Study to Investigate the Safety, Tolerability, and Pharmacokinetics of CCI15106 Inhalation Powder in Healthy Participants and Participants With Moderate Chronic Obstructive Pulmonary Disease (COPD) Including Evaluation of Environmental and Healthy By-stander Exposure Levels During Dosing
Brief Title: Study of Safety and Drug Levels of CCI15106 Inhalation Powder in Healthy Adults and Adults With Moderate Chronic Obstructive Pulmonary Disease. Study of CCI15106 Levels in People Standing Near the Person Inhaling the Drug
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205822; 2017-001070-42 (EudraCT Number)
Record Dates: First submitted 2017-07-11; First posted 2017-08-01 (Actual); Results first posted 2019-09-27 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: bystander; inhalation powder; monodose device; COPD; pharmacokinetics; safety; Healthy; CCI15106; tolerability
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: In this study, subjects will be randomized to receive either study drug or placebo in a parallel manner.
Who Masked: Participant, Investigator
Masking Description: This is a double blind, randomized study and subject and investigator will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Cohort A, Part 1: Active (Experimental): 60 milligrams (mg) single dose of CCI15106 will be administered by inhalation route on Day 1; 120 mg single dose will be administered on Day 3; and then 30 mg dose will be administered twice daily (BID) on Days 6-19 to healthy subjects.
  Interventions: Drug: CCI15106
- Cohort A, Part 1: Placebo (Placebo Comparator): 60 mg single dose of placebo will be administered by inhalation route on Day 1; 120 mg single dose will be administered on Day 3; and then 30 mg dose will be administered BID on Days 6-19 to healthy subjects.
  Interventions: Drug: Placebo
- Cohort B, Part 1: Active (Experimental): 60 mg of CCI15106 BID will be administered by inhalation route for 14 days to healthy subjects.
  Interventions: Drug: CCI15106
- Cohort B, Part 1: Placebo (Placebo Comparator): 60 mg of placebo BID will be administered by inhalation route for 14 days to healthy subjects.
  Interventions: Drug: Placebo
- Cohort C, Part 1: bystanders (No Intervention): Healthy subjects will be enrolled to follow bystander exposure and will be studied concomitantly with Cohort B.
- Cohort A, Part 2: Active (Experimental): 60 mg single dose of CCI15106 will be administered by inhalation route to subjects with COPD.
  Interventions: Drug: CCI15106
- Cohort A, Part 2: Placebo (Placebo Comparator): 60 mg single dose of placebo will be administered by inhalation route to subjects with COPD.
  Interventions: Drug: Placebo
- Cohort B, Part 2: Active (Experimental): 60 mg BID dose of CCI15106 will be administered by inhalation route for 14 days to subjects with COPD.
  Interventions: Drug: CCI15106
- Cohort B, Part 2: Placebo (Placebo Comparator): 60 mg BID dose of placebo will be administered by inhalation route for 14 days to subjects with COPD.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CCI15106 — One capsule (single dose or repeat dose) of 30 mg of CCI15106 will be administered to healthy subjects and subjects with COPD via inhalation route using Monodose RS01 device. The morning dose will be taken in fasting state and for repeat dose; the evening dose will be taken at least 2 hours after food.
  Arms: Cohort A, Part 1: Active; Cohort A, Part 2: Active; Cohort B, Part 1: Active; Cohort B, Part 2: Active
Drug: Placebo — One capsule of placebo will be administered to healthy subjects and subjects with COPD via inhalation route using Monodose RS01 device. The morning dose will be taken in fasting state and for repeat dose; the evening dose will be taken at least 2 hours after food.
  Arms: Cohort A, Part 1: Placebo; Cohort A, Part 2: Placebo; Cohort B, Part 1: Placebo; Cohort B, Part 2: Placebo

SUMMARY:
This single and repeat increasing dose study will collect information on safety, tolerability and drug levels in the body of the CCI15106 inhalation powder. The study will also look at the level of CCI15106 that will be released into the air and may be found in the blood of the people standing around the person inhaling it (bystanders). This is a two-part study in which Part 1 will enroll healthy subjects and look at environmental and bystander exposure and Part 2 will enroll subjects with moderate COPD. Approximately 36 healthy subjects and approximately 22 subjects with COPD will be randomized in this study for dosing. The total study duration will be 82 days for Cohort A Part 1; 75 days for Cohort B Part 1 and Cohort C Part 1; 77 days for Cohort A Part 2; and 90 days for Cohort B Part 2.

ELIGIBILITY:
Some important Inclusion Criteria:

For healthy subjects and bystanders:

* 18 to 65 years of age.
* Healthy as determined by a doctor.
* Men who agree to use contraception during the treatment period and for at least 7 months after the last dose of study medicine and agree not to donate sperm during this period.
* Women who are not pregnant or breastfeeding, and not of childbearing potential.

For subjects with COPD:

* 40 to 75 years of age.
* Diagnosed with moderate COPD by a doctor.
* Have breathing test results that are consistent with moderate COPD as defined in the study protocol.
* A smoker or an ex-smoker.
* Men who agree to use contraception during the treatment period and for at least 7 months after the last dose of study medicine and agree not to donate sperm during this period.
* Women who are not pregnant or breastfeeding, and not of childbearing potential.

Some Important Exclusion Criteria:

For healthy subjects and bystanders:

* History of liver disease.
* Use of over-the-counter or prescription drugs (including vitamins) 7 days before the study until completion of the follow-up visit.
* Participation in the study would result in loss of more than 500 milliliter (mL) of blood within 3 months.
* Participation in another clinical trial with an investigational product within about 3 months before this study.
* Positive drug/alcohol screen.
* Regular use of known drugs of abuse.
* Regular alcohol consumption within 3 months before the study.
* Breath test indicative of smoking at study start.
* Documented lactose allergy/intolerance.
* Men whose partner is pregnant or breastfeeding cannot participate.
* Certain blood test results may not allow subjects to participate, as described in the study protocol.

For subjects with COPD:

* History of liver disease.
* Poorly controlled COPD disease as, for example, more than 2 exacerbations of COPD per year.
* Some respiratory conditions, like for example active tuberculosis, lung cancer or any other respiratory condition. Subjects with other respiratory conditions (for example, clinically significant: asthma, pulmonary fibrosis, bronchiectasis) are excluded if these conditions are the primary cause of their respiratory symptoms.
* Unstable or uncontrolled cardiac disease.
* Problems with kidney function as defined in the study protocol.
* Past or current medical conditions or diseases that are not well controlled.
* Subjects are not allowed to take oral corticosteroids from 4 weeks prior to screening and for the duration of the study.
* Subjects taking medications for any chronic conditions have to be on stable doses for 4 weeks before screening and until after study treatment is finished.
* Use of short-acting inhaled bronchodilators is allowed, but subjects must be able to stop their medications several times during the study.
* Use of long-acting bronchodilators is allowed, but subjects must be able to change the schedule of their medications twice during the study.
* Participation in the study would result in loss of more than 500 mL within 3 months.
* Participation in another clinical trial with an investigational product within about 3 months before this study.
* Positive drug/alcohol screen.
* Regular use of known drugs of abuse.
* Regular alcohol consumption within 3 months before the study.
* Unable to refrain from smoking for certain periods during the study (maximum about 6 hours).
* Documented lactose allergy/intolerance.
* Men whose partner is pregnant or breastfeeding cannot participate.
* Certain blood test results may not allow subjects to participate, as described in the study protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-07-13 (Actual); Primary Completion 2018-06-19 (Actual); Study Completion 2018-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Park Royal, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20373

REFERENCES:
- [Derived] Dumont EF, Oliver AJ, Ioannou C, Billiard J, Dennison J, van den Berg F, Yang S, Chandrasekaran V, Young GC, Lahiry A, Starbuck DC, Harrell AW, Georgiou A, Hopchet N, Gillies A, Baker SJ. A Novel Inhaled Dry-Powder Formulation of Ribavirin Allows for Efficient Lung Delivery in Healthy Participants and Those with Chronic Obstructive Pulmonary Disease in a Phase 1 Study. Antimicrob Agents Chemother. 2020 Apr 21;64(5):e02267-19. doi: 10.1128/AAC.02267-19. Print 2020 Apr 21. PMID 32071044

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a two parts single and repeat dose escalation study. Part 1 was conducted in healthy volunteers and Part 2 was conducted in participants with moderate chronic obstructive pulmonary disease (COPD).
Pre-assignment Details: A total of 52 participants (36 in Part 1 and 16 in Part 2) were enrolled in this study. This study was conducted at a single center in the United Kingdom from 13-July-2017 to 19-June-2018.
Groups:
- Part 1: Cohort A- CCI15106 60 mg SD: Healthy participants were administered a single dose (SD) of CCI15106 60 mg by inhalation route on Day 1 via Monodose RS01.
- Part 1: Cohort A- CCI15106 120 mg SD: Healthy participants were administered a SD of CCI15106 120 mg by inhalation route on Day 3 via Monodose RS01.
- Part 1: Cohort A- CCI15106 30 mg BID: Healthy participants were administered a twice daily (BID) dose of CCI15106 30 mg by inhalation route on Days 6 to 19 via Monodose RS01.
- Part 1: Cohort A- Placebo: Healthy participants were administered a SD of matching placebo 60 mg by inhalation route on Day 1 via Monodose RS01; followed by a SD matching placebo 120 mg by inhalation route on Day 3 via Monodose RS01; further followed by a BID dose of matching placebo 30 mg by inhalation route on Days 6 to 19 via Monodose RS01 in cohort A.
- Part 1: Cohort B- CCI15106 60 mg BID: Healthy participants were administered with a BID dose of CCI15106 60 mg by inhalation route on Days 1 to 14 via Monodose RS01.
- Part 1: Cohort B- Placebo: Healthy participants were administered with a BID dose of matching placebo 60 mg by inhalation route on Days 1 to 14 via Monodose RS01 in cohort B.
- Part 1: Cohort C- Bystanders: Healthy participants were enrolled to evaluate bystander exposure and evaluated concomitantly with Cohort B. Bystanders reported to the unit on Day -1 and remained for 14 days of dosing of Cohort B.
- Part 2: Cohort A- CCI15106 60 mg SD: Participants with COPD received a SD of CCI15106 60 mg by inhalation route on Day 1 via Monodose RS01.
- Part 2: Cohort A- Placebo: Participants with COPD received a SD of matching placebo 60 mg by inhalation route on Day 1 via Monodose RS01 in Cohort A.
- Part 2: Cohort B- CCI15106 60 mg BID: Participants with COPD received a BID of CCI15106 60 mg by inhalation route on Days 1 to 14 via Monodose RS01.
Period: Part 1 (Cohort A 60 mg - Day 1)
Arm/Group | Part 1: Cohort A- CCI15106 60 mg SD | Part 1: Cohort A- CCI15106 120 mg SD | Part 1: Cohort A- CCI15106 30 mg BID | Part 1: Cohort A- Placebo | Part 1: Cohort B- CCI15106 60 mg BID | Part 1: Cohort B- Placebo | Part 1: Cohort C- Bystanders | Part 2: Cohort A- CCI15106 60 mg SD | Part 2: Cohort A- Placebo | Part 2: Cohort B- CCI15106 60 mg BID
Started | 6 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 6 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1 (Cohort A 120 mg - Day 3)
Arm/Group | Part 1: Cohort A- CCI15106 60 mg SD | Part 1: Cohort A- CCI15106 120 mg SD | Part 1: Cohort A- CCI15106 30 mg BID | Part 1: Cohort A- Placebo | Part 1: Cohort B- CCI15106 60 mg BID | Part 1: Cohort B- Placebo | Part 1: Cohort C- Bystanders | Part 2: Cohort A- CCI15106 60 mg SD | Part 2: Cohort A- Placebo | Part 2: Cohort B- CCI15106 60 mg BID
Started | 0 | 6 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 6 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1 (Cohort A 30mg BID-Days 6 to 19)
Arm/Group | Part 1: Cohort A- CCI15106 60 mg SD | Part 1: Cohort A- CCI15106 120 mg SD | Part 1: Cohort A- CCI15106 30 mg BID | Part 1: Cohort A- Placebo | Part 1: Cohort B- CCI15106 60 mg BID | Part 1: Cohort B- Placebo | Part 1: Cohort C- Bystanders | Part 2: Cohort A- CCI15106 60 mg SD | Part 2: Cohort A- Placebo | Part 2: Cohort B- CCI15106 60 mg BID
Started | 0 | 0 | 6 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 6 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1 (Cohort B and C- Days 1 to 14)
Arm/Group | Part 1: Cohort A- CCI15106 60 mg SD | Part 1: Cohort A- CCI15106 120 mg SD | Part 1: Cohort A- CCI15106 30 mg BID | Part 1: Cohort A- Placebo | Part 1: Cohort B- CCI15106 60 mg BID | Part 1: Cohort B- Placebo | Part 1: Cohort C- Bystanders | Part 2: Cohort A- CCI15106 60 mg SD | Part 2: Cohort A- Placebo | Part 2: Cohort B- CCI15106 60 mg BID
Started | 0 | 0 | 0 | 0 | 12 | 2 | 14 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 10 | 2 | 14 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Drug was prematurely discontinued | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Part 2 (Cohort A - Day 1)
Arm/Group | Part 1: Cohort A- CCI15106 60 mg SD | Part 1: Cohort A- CCI15106 120 mg SD | Part 1: Cohort A- CCI15106 30 mg BID | Part 1: Cohort A- Placebo | Part 1: Cohort B- CCI15106 60 mg BID | Part 1: Cohort B- Placebo | Part 1: Cohort C- Bystanders | Part 2: Cohort A- CCI15106 60 mg SD | Part 2: Cohort A- Placebo | Part 2: Cohort B- CCI15106 60 mg BID
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2 (Cohort B - Days 1 to 14)
Arm/Group | Part 1: Cohort A- CCI15106 60 mg SD | Part 1: Cohort A- CCI15106 120 mg SD | Part 1: Cohort A- CCI15106 30 mg BID | Part 1: Cohort A- Placebo | Part 1: Cohort B- CCI15106 60 mg BID | Part 1: Cohort B- Placebo | Part 1: Cohort C- Bystanders | Part 2: Cohort A- CCI15106 60 mg SD | Part 2: Cohort A- Placebo | Part 2: Cohort B- CCI15106 60 mg BID
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 1: Cohort A- CCI15106: Healthy participants were administered a SD dose of CCI15106 60 mg by inhalation route on Day 1 via Monodose RS01, followed by a SD dose of CCI15106 120 mg by inhalation route on Day 3 via Monodose RS01, further followed by a BID dose of CCI15106 30 mg by inhalation route on Days 6 to 19 via Monodose RS01.
- Part 1: Cohort A- Placebo: Healthy participants were administered a SD dose of matching placebo 60 mg by inhalation route on Day 1 via Monodose RS01, followed by a SD dose of matching placebo 120 mg by inhalation route on Day 3 via Monodose RS01, further followed by a BID dose of matching placebo 30 mg by inhalation route on Days 6 to 19 via Monodose RS01.
- Total: Total of all reporting groups
Arm/Group | Part 1: Cohort A- CCI15106 | Part 1: Cohort A- Placebo | Part 1: Cohort B- CCI15106 60 mg BID | Part 1: Cohort B- Placebo | Part 1: Cohort C- Bystanders | Part 2: Cohort A- CCI15106 60 mg SD | Part 2: Cohort A- Placebo | Part 2: Cohort B- CCI15106 60 mg BID | Total
Number analyzed (Participants) | 6 | 2 | 12 | 2 | 14 | 6 | 2 | 8 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 2 | 12 | 2 | 14 | 4 | 1 | 4 | 45
  >=65 years | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 4 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 5
  Male | 6 | 2 | 12 | 2 | 13 | 4 | 2 | 6 | 47
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 6
  White-White/Caucasian/European | 5 | 2 | 10 | 1 | 9 | 6 | 2 | 8 | 43
  Black or African American and White | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
  Black or African American and Asian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Part 1 Cohort A: Number of Participants With Non-serious Adverse Events (NSAEs) and Serious Adverse Events (SAEs) in CCI15106
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. An SAE is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other situations judged by physician. Safety population comprised of all participants who received at least one dose of study treatment during the study.
Time Frame: Up to 51 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Cohort A- CCI15106 60 mg SD: Healthy participants were administered a SD of CCI15106 60 mg by inhalation route on Day 1 via Monodose RS01.
- Part 1: Cohort A- CCI15106 30 mg BID: Healthy participants were administered a BID dose of CCI15106 30 mg by inhalation route on Days 6 to 19 via Monodose RS01.
Arm/Group | Part 1: Cohort A- CCI15106 60 mg SD | Part 1: Cohort A- CCI15106 120 mg SD | Part 1: Cohort A- CCI15106 30 mg BID | Part 1: Cohort A- Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 2
Participants
  NSAEs | 0 | 0 | 0 | 0
  SAEs | 0 | 0 | 0 | 0

2. Primary Outcome: Part 1 Cohort B: Number of Participants With NSAEs and SAEs in CCI15106
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. An SAE is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other situations judged by physician.
Time Frame: Up to 46 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort B- CCI15106 60 mg BID | Part 1: Cohort B- Placebo
Number analyzed (Participants) | 12 | 2
Participants
  NSAEs | 6 | 0
  SAEs | 0 | 0

3. Primary Outcome: Part 1 Cohort C: Number of Participants With NSAEs and SAEs in Bystanders
Description: as for outcome 2
Time Frame: Up to 46 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort C- Bystanders
Number analyzed (Participants) | 14
Participants
  NSAEs | 6
  SAEs | 0

4. Primary Outcome: Part 2 Cohort A: Number of Participants With NSAEs and SAEs
Description: as for outcome 2
Time Frame: Up to 33 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Cohort A- CCI15106 60 mg SD | Part 2: Cohort A- Placebo
Number analyzed (Participants) | 6 | 2
Participants
  NSAEs | 0 | 0
  SAEs | 0 | 0

5. Primary Outcome: Part 2 Cohort B: Number of Participants With NSAEs and SAEs
Description: as for outcome 2
Time Frame: Up to 46 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Cohort B- CCI15106 60 mg BID
Number analyzed (Participants) | 8
Participants
  NSAEs | 7
  SAEs | 0

6. Primary Outcome: Part 1: Number of Participants With Hematology Values of Potential Clinical Importance (PCI) in CCI15106
Description: PCI ranges for the hematology parameters were as follows: hematocrit (high: >0.54 proportion of red blood cell [RBC] in blood for male, >0.54 proportion of RBC in blood for female), hemoglobin (high: >180 grams [g]/L in male, >180 g/L in female), lymphocytes (low: <0.8 10^9/L), neutrophil count (low: <1.5 10^9/L) and platelet count (low: <100 10^9/L and high: 550 10^9/L). Data for the participants with high and low values has been reported.
Time Frame: Up to 51 days
Population: Safety Population. The primary aim was to compare the safety profiles of the different active doses; hence, placebo arms have been combined as pre-specified in reporting and analysis plan.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Placebo: Healthy participants were administered a SD of matching placebo 60 mg by inhalation route on Day 1 via Monodose RS01; followed by a SD matching placebo 120 mg by inhalation route on Day 3 via Monodose RS01; followed by a BID dose of matching placebo 30 mg by inhalation route on Days 6 to 19 via Monodose RS01 in cohort A; further followed by a BID dose of CCI15106 60 mg by inhalation route on Days 1 to 14 via Monodose RS01 in cohort B.
Arm/Group | Part 1: Cohort A- CCI15106 60 mg SD | Part 1: Cohort A- CCI15106 120 mg SD | Part 1: Cohort A- CCI15106 30 mg BID | Part 1: Cohort B- CCI15106 60 mg BID | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 12 | 4
Participants
  Hematocrit: high | 0 | 0 | 0 | 0 | 0
  Hemoglobin: high | 0 | 0 | 0 | 0 | 0
  Lymphocytes: low | 0 | 0 | 0 | 0 | 0
  Neutrophil count: low | 0 | 1 | 0 | 0 | 0
  Platelet count: low | 0 | 0 | 0 | 0 | 0
  Platelet count: high | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Part 1: Number of Participants With Hematology Values of PCI in Bystanders
Description: PCI ranges for the hematology parameters were as follows: hematocrit (high: >0.54 proportion of RBC in blood for male, >0.54 proportion of RBC in blood for female), hemoglobin (high: >180 g/L in male, >180 g/L in female), lymphocytes (low: <0.8 10^9/L), neutrophil count (low: <1.5 10^9/L) and platelet count (low: <100 10^9/L and high: 550 10^9/L). Data for the participants with high and low values has been reported.
Time Frame: Up to 46 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort C- Bystanders
Number analyzed (Participants) | 14
Participants
  Hematocrit: high | 0
  Hemoglobin: high | 0
  Lymphocytes: low | 0
  Neutrophil count: low | 0
  Platelet count: low | 0
  Platelet count: high | 0

8. Primary Outcome: Part 2: Number of Participants With Hematology Values of PCI
Description: as for outcome 7
Time Frame: Up to 46 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Cohort A- CCI15106 60 mg SD | Part 2: Cohort A- Placebo | Part 2: Cohort B- CCI15106 60 mg BID
Number analyzed (Participants) | 6 | 2 | 8
Participants
  Hematocrit: high | 0 | 0 | 0
  Hemoglobin: high | 0 | 0 | 0
  Lymphocytes: low | 0 | 0 | 0
  Neutrophil count: low | 0 | 0 | 0
  Platelet count: low | 0 | 0 | 0
  Platelet count: high | 0 | 0 | 0

9. Primary Outcome: Part 1: Number of Participants With Clinical Chemistry Values of PCI in CCI15106
Description: PCI ranges for the clinical chemistry parameters were as follows: albumin (low: <30 millimole per liter [mmol/L]), calcium (low: <2 mmol/L and high: >2.75 mmol/L), glucose (low: <3 mmol/L and high: >9 mmol/L), potassium (low: <3 mmol/L and high: >5.5 mmol/L) and sodium (low: <130 mmol/L and high: >150 mmol/L). Data for the participants with high and low values has been reported.
Time Frame: Up to 51 days
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort A- CCI15106 60 mg SD | Part 1: Cohort A- CCI15106 120 mg SD | Part 1: Cohort A- CCI15106 30 mg BID | Part 1: Cohort B- CCI15106 60 mg BID | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 12 | 4
Participants
  Albumin: low | 0 | 0 | 0 | 0 | 0
  Calcium: low | 0 | 0 | 0 | 0 | 0
  Calcium: high | 0 | 0 | 0 | 0 | 0
  Glucose: low | 0 | 0 | 0 | 0 | 0
  Glucose: high | 0 | 0 | 0 | 0 | 0
  Potassium: low | 0 | 0 | 0 | 0 | 0
  Potassium: high | 0 | 0 | 0 | 0 | 0
  Sodium: low | 0 | 0 | 0 | 0 | 0
  Sodium: high | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Part 1: Number of Participants With Clinical Chemistry Values of PCI in Bystanders
Description: PCI ranges for the clinical chemistry parameters were as follows: albumin (low: <30 mmol/L), calcium (low: <2 mmol/L and high: >2.75 mmol/L), glucose (low: <3 mmol/L and high: >9 mmol/L), potassium (low: <3 mmol/L and high: >5.5 mmol/L) and sodium (low: <130 mmol/L and high: >150 mmol/L). Data for the participants with high and low values has been reported.
Time Frame: Up to 46 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort C- Bystanders
Number analyzed (Participants) | 14
Participants
  Albumin: low | 0
  Calcium: low | 0
  Calcium: high | 0
  Glucose: low | 0
  Glucose: high | 0
  Potassium: low | 0
  Potassium: high | 0
  Sodium: low | 0
  Sodium: high | 0

11. Primary Outcome: Part 2: Number of Participants With Clinical Chemistry Values of PCI
Description: as for outcome 10
Time Frame: Up to 46 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Cohort A- CCI15106 60 mg SD | Part 2: Cohort A- Placebo | Part 2: Cohort B- CCI15106 60 mg BID
Number analyzed (Participants) | 6 | 2 | 8
Participants
  Albumin: low | 0 | 0 | 0
  Calcium: low | 0 | 0 | 0
  Calcium: high | 0 | 0 | 0
  Glucose: low | 0 | 0 | 0
  Glucose: high | 0 | 0 | 1
  Potassium: low | 0 | 0 | 0
  Potassium: high | 0 | 0 | 0
  Sodium: low | 0 | 0 | 0
  Sodium: high | 0 | 0 | 0

12. Primary Outcome: Part 1 Cohort A: Potential of Hydrogen (pH) Value by Visit- CCI15106 60 mg SD
Description: Urine samples were collected from participants at indicated time points for analysis of pH. Baseline was considered as the latest pre-dose assessment with a non-missing value for Baseline (Day -1).
Time Frame: Baseline (Day -1) and Day 2
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part 1: Cohort A- CCI15106 60 mg SD
Number analyzed (Participants) | 6
pH
  Baseline | 6.00 (0.000)
  Day 2 | 6.33 (0.816)

13. Primary Outcome: Part 1 Cohort A: pH Value by Visit- CCI15106 120 mg SD
Description: Urine sample was collected from participants at indicated time point for analysis of pH.
Time Frame: Day 5
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part 1: Cohort A- CCI15106 120 mg SD
Number analyzed (Participants) | 6
pH | 6.58 (0.736)

14. Primary Outcome: Part 1 Cohort A: pH Value by Visit- CCI15106 30 mg BID
Description: Urine samples were collected from participants at indicated time points for analysis of pH.
Time Frame: Days 12 and 22
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part 1: Cohort A- CCI15106 30 mg BID
Number analyzed (Participants) | 6
pH
  Day 12 | 6.50 (0.949)
  Day 22 | 6.92 (0.665)

15. Primary Outcome: Part 1 Cohort B: pH Value by Visit- CCI15106 60 mg BID
Description: as for outcome 12
Time Frame: Baseline (Day -1), Days 7 and 15
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part 1: Cohort B- CCI15106 60 mg BID
Number analyzed (Participants) | 12
pH
  Baseline | 6.21 (0.811)
  Day 7 | 6.63 (0.882)
  Day 15 | 6.21 (0.620)

16. Primary Outcome: Part 1: pH Value by Visit- Placebo
Description: as for outcome 12
Time Frame: Baseline (Day -1), Days 2, 5, 7, 12, 15 and 22
Population: Safety Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). The primary aim was to compare the safety profiles of the different active doses; hence, placebo arms have been combined as pre-specified in reporting and analysis plan.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part 1: Placebo
Number analyzed (Participants) | 4
pH
  Baseline: n=4 | 6.50 (0.707)
  Day 2: n=2: number analyzed (Participants) | 2
  Day 2: n=2 | 5.50 (0.707)
  Day 5: n=2: number analyzed (Participants) | 2
  Day 5: n=2 | 6.25 (0.354)
  Day 7: n=2: number analyzed (Participants) | 2
  Day 7: n=2 | 7.00 (1.414)
  Day 12: n=2: number analyzed (Participants) | 2
  Day 12: n=2 | 5.75 (1.061)
  Day 15: n=2: number analyzed (Participants) | 2
  Day 15: n=2 | 5.50 (0.707)
  Day 22: n=2: number analyzed (Participants) | 2
  Day 22: n=2 | 6.75 (1.061)

17. Primary Outcome: Part 1 Cohort C: pH Value by Visit- CCI15106 in Bystanders
Description: as for outcome 12
Time Frame: Baseline (Day -1), Days 7 and 15
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part 1: Cohort C- Bystanders
Number analyzed (Participants) | 14
pH
  Baseline | 6.36 (0.633)
  Day 7 | 6.36 (0.719)
  Day 15 | 5.96 (0.499)

18. Primary Outcome: Part 2 Cohort A: pH Value by Visit- CCI15106
Description: as for outcome 12
Time Frame: Baseline (Day -1) and Day 2
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part 2: Cohort A- CCI15106 60 mg SD | Part 2: Cohort A- Placebo
Number analyzed (Participants) | 6 | 2
pH
  Baseline | 6.25 (0.822) | 6.75 (1.061)
  Day 2 | 6.58 (0.801) | 6.50 (0.707)

19. Primary Outcome: Part 2 Cohort B: pH Value by Visit- CCI15106 60 mg BID
Description: as for outcome 12
Time Frame: Baseline (Day -1), Days 7 and 15
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part 2: Cohort B- CCI15106 60 mg BID
Number analyzed (Participants) | 8
pH
  Baseline | 6.13 (0.916)
  Day 7 | 5.94 (0.863)
  Day 15 | 5.81 (0.884)

20. Primary Outcome: Part 1 Cohort A: Specific Gravity Value by Visit- CCI15106 60 mg SD
Description: Urinary specific gravity measurement is a routine part of urinalysis. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. The concentration of the excreted molecules determines the urine's specific gravity. Urine samples were collected from participants at indicated time points for analysis of specific gravity. Baseline was considered as the latest pre-dose assessment with a non-missing value for Baseline (Day -1).
Time Frame: Baseline (Day -1) and Day 2
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 1: Cohort A- CCI15106 60 mg SD
Number analyzed (Participants) | 6
Ratio
  Baseline | 1.0217 (0.01033)
  Day 2 | 1.0105 (0.00625)

21. Primary Outcome: Part 1 Cohort A: Specific Gravity Value by Visit- CCI15106 120 mg SD
Description: Urinary specific gravity measurement is a routine part of urinalysis. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. The concentration of the excreted molecules determines the urine's specific gravity. Urine sample was collected from participants at indicated time point for analysis of specific gravity.
Time Frame: Day 5
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 1: Cohort A- CCI15106 120 mg SD
Number analyzed (Participants) | 6
Ratio | 1.0182 (0.00722)

22. Primary Outcome: Part 1 Cohort A: Specific Gravity Value by Visit- CCI15106 30 mg BID
Description: Urinary specific gravity measurement is a routine part of urinalysis. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. The concentration of the excreted molecules determines the urine's specific gravity. Urine samples were collected from participants at indicated time points for analysis of specific gravity.
Time Frame: Days 12 and 22
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 1: Cohort A- CCI15106 30 mg BID
Number analyzed (Participants) | 6
Ratio
  Day 12 | 1.0115 (0.00442)
  Day 22 | 1.0115 (0.00442)

23. Primary Outcome: Part 1 Cohort B: Specific Gravity Value by Visit- CCI15106 60 mg BID
Description: as for outcome 20
Time Frame: Baseline (Day -1), Days 7 and 15
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 1: Cohort B- CCI15106 60 mg BID
Number analyzed (Participants) | 12
Ratio
  Baseline | 1.0136 (0.00734)
  Day 7 | 1.0152 (0.01039)
  Day 15 | 1.0167 (0.00444)

24. Primary Outcome: Part 1: Specific Gravity Value by Visit- Placebo
Description: as for outcome 20
Time Frame: Baseline (Day -1), Days 2, 5, 7, 12, 15 and 22
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 1: Placebo
Number analyzed (Participants) | 4
Ratio
  Baseline: n=4 | 1.0148 (0.00858)
  Day 2: n=2: number analyzed (Participants) | 2
  Day 2: n=2 | 1.0150 (0.00000)
  Day 5: n=2: number analyzed (Participants) | 2
  Day 5: n=2 | 1.0150 (0.00707)
  Day 7: n=2: number analyzed (Participants) | 2
  Day 7: n=2 | 1.0150 (0.00707)
  Day 12: n=2: number analyzed (Participants) | 2
  Day 12: n=2 | 1.0120 (0.01131)
  Day 15: n=2: number analyzed (Participants) | 2
  Day 15: n=2 | 1.0150 (0.00707)
  Day 22: n=2: number analyzed (Participants) | 2
  Day 22: n=2 | 1.0095 (0.00778)

25. Primary Outcome: Part 1 Cohort C: Specific Gravity Value by Visit- CCI15106 in Bystanders
Description: as for outcome 20
Time Frame: Baseline (Day -1), Days 7 and 15
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 1: Cohort C- Bystanders
Number analyzed (Participants) | 14
Ratio
  Baseline | 1.0191 (0.01339)
  Day 7 | 1.0163 (0.00907)
  Day 15 | 1.0182 (0.00750)

26. Primary Outcome: Part 2 Cohort A: Specific Gravity Value by Visit- CCI15106
Description: as for outcome 20
Time Frame: Baseline (Day -1) and Day 2
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 2: Cohort A- CCI15106 60 mg SD | Part 2: Cohort A- Placebo
Number analyzed (Participants) | 6 | 2
Ratio
  Baseline | 1.0205 (0.01694) | 1.0175 (0.01061)
  Day 2 | 1.0147 (0.00737) | 1.0275 (0.01768)

27. Primary Outcome: Part 2 Cohort B: Specific Gravity Value by Visit- CCI15106 60 mg BID
Description: as for outcome 20
Time Frame: Baseline (Day -1), Days 7 and 15
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 2: Cohort B- CCI15106 60 mg BID
Number analyzed (Participants) | 8
Ratio
  Baseline | 1.0106 (0.00678)
  Day 7 | 1.0114 (0.00424)
  Day 15 | 1.0133 (0.00523)

28. Primary Outcome: Part 1: Number of Participants With Worst Case Post-Baseline 12-lead Electrocardiogram (ECG) of PCI in CCI15106
Description: PCI ranges for the ECG parameters were as follows: absolute QTc interval >450 and <480, >=480 and <500, >=500 milliseconds (msec), absolute PR interval <110 and >220 msec and absolute QRS interval <75 and >110 msec. QTcF=Frederica's QT interval corrected for heart rate; QTcB=Bazett's QT interval corrected for heart rate. Data for worst case post-Baseline has been reported.
Time Frame: Up to 51 days
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort A- CCI15106 60 mg SD | Part 1: Cohort A- CCI15106 120 mg SD | Part 1: Cohort A- CCI15106 30 mg BID | Part 1: Cohort B- CCI15106 60 mg BID | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 12 | 4
Participants
  PR interval: Value<110 | 0 | 0 | 0 | 0 | 0
  PR interval: 110<=Value<=220 | 6 | 6 | 6 | 12 | 4
  PR interval: Value>220 | 0 | 0 | 0 | 0 | 0
  QRS duration: Value<75 | 0 | 0 | 0 | 0 | 0
  QRS duration: 75<=Value<=110 | 4 | 6 | 5 | 9 | 3
  QRS duration: Value>110 | 2 | 0 | 1 | 3 | 1
  QT interval: Value<=450 | 5 | 6 | 6 | 11 | 4
  QT interval: 450<Value<480 | 1 | 0 | 0 | 1 | 0
  QT interval: 480<=Value<500 | 0 | 0 | 0 | 0 | 0
  QT interval: Value>=500 | 0 | 0 | 0 | 0 | 0
  QTcB interval: Value<=450 | 6 | 6 | 6 | 8 | 4
  QTcB interval: 450<Value<480 | 0 | 0 | 0 | 4 | 0
  QTcB interval: 480<=Value<500 | 0 | 0 | 0 | 0 | 0
  QTcB interval: Value>=500 | 0 | 0 | 0 | 0 | 0
  QTcF interval: Value<=450 | 6 | 6 | 6 | 11 | 4
  QTcF interval: 450<Value<480 | 0 | 0 | 0 | 1 | 0
  QTcF interval: 480<=Value<500 | 0 | 0 | 0 | 0 | 0
  QTcF interval: Value>=500 | 0 | 0 | 0 | 0 | 0

29. Primary Outcome: Part 1: Number of Participants With Worst Case Post-Baseline 12-lead ECG of PCI in Bystander
Description: PCI ranges for the ECG parameters were as follows: absolute QTc interval >450 and <480, >=480 and <500, >=500 msec, absolute PR interval <110 and >220 msec and absolute QRS interval <75 and >110 msec. Data for worst case post-Baseline has been reported.
Time Frame: Up to 46 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort C- Bystanders
Number analyzed (Participants) | 14
Participants
  PR interval: Value<110 | 0
  PR interval: 110<=Value<=220 | 14
  PR interval: Value>220 | 0
  QRS duration: Value<75 | 0
  QRS duration: 75<=Value<=110 | 13
  QRS duration: Value>110 | 1
  QT interval: Value<=450 | 13
  QT interval: 450<Value<480 | 1
  QT interval: 480<=Value<500 | 0
  QT interval: Value>=500 | 0
  QTcB interval: Value<=450 | 14
  QTcB interval: 450<Value<480 | 0
  QTcB interval: 480<=Value<500 | 0
  QTcB interval: Value>=500 | 0
  QTcF interval: Value<=450 | 14
  QTcF interval: 450<Value<480 | 0
  QTcF interval: 480<=Value<500 | 0
  QTcF interval: Value>=500 | 0

30. Primary Outcome: Part 2: Number of Participants With Worst Case Post-Baseline 12-lead ECG of PCI
Description: as for outcome 29
Time Frame: Up to 46 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Cohort A- CCI15106 60 mg SD | Part 2: Cohort A- Placebo | Part 2: Cohort B- CCI15106 60 mg BID
Number analyzed (Participants) | 6 | 2 | 8
Participants
  PR interval: Value<110 | 1 | 0 | 0
  PR interval: 110<=Value<=220 | 5 | 2 | 8
  PR interval: Value>220 | 0 | 0 | 0
  QRS duration: Value<75 | 1 | 0 | 0
  QRS duration: 75<=Value<=110 | 5 | 2 | 7
  QRS duration: Value>110 | 0 | 0 | 1
  QT interval: Value<=450 | 6 | 2 | 8
  QT interval: 450<Value<480 | 0 | 0 | 0
  QT interval: 480<=Value<500 | 0 | 0 | 0
  QT interval: Value>=500 | 0 | 0 | 0
  QTcB interval: Value<=450 | 5 | 2 | 7
  QTcB interval: 450<Value<480 | 1 | 0 | 1
  QTcB interval: 480<=Value<500 | 0 | 0 | 0
  QTcB interval: Value>=500 | 0 | 0 | 0
  QTcF interval: Value<=450 | 6 | 2 | 7
  QTcF interval: 450<Value<480 | 0 | 0 | 1
  QTcF interval: 480<=Value<500 | 0 | 0 | 0
  QTcF interval: Value>=500 | 0 | 0 | 0

31. Primary Outcome: Part 1: Number of Participants With Abnormal Telemetry Findings
Description: Continuous cardiac telemetry was performed from approximately 0.5 hour (pre-dose) to 4 hours post-dose. Abnormal findings were categorized as clinically significant (CS) and not clinically significant (NCS). Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: Days 1, 3, 6, 7, 12 and 18: 0.5 hour (pre-dose) to 4 hours post-dose
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort A- CCI15106 60 mg SD | Part 1: Cohort A- CCI15106 120 mg SD | Part 1: Cohort A- CCI15106 30 mg BID | Part 1: Cohort B- CCI15106 60 mg BID | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 12 | 4
Participants
  Day 1: 0.5 to 4 hours post-dose-CS;n=6,0,0,12,4: number analyzed (Participants) | 6 | 0 | 0 | 12 | 4
  Day 1: 0.5 to 4 hours post-dose-CS;n=6,0,0,12,4 | 0 |  |  | 0 | 0
  Day 1: 0.5 to 4 hours post-dose-NCS;n=6,0,0,12,4: number analyzed (Participants) | 6 | 0 | 0 | 12 | 4
  Day 1: 0.5 to 4 hours post-dose-NCS;n=6,0,0,12,4 | 0 |  |  | 0 | 0
  Day 3: 0.5 to 4 hours post-dose-CS;n=0,6,0,0,2: number analyzed (Participants) | 0 | 6 | 0 | 0 | 2
  Day 3: 0.5 to 4 hours post-dose-CS;n=0,6,0,0,2 |  | 0 |  |  | 0
  Day 3: 0.5 to 4 hours post-dose-NCS;n=0,6,0,0,2: number analyzed (Participants) | 0 | 6 | 0 | 0 | 2
  Day 3: 0.5 to 4 hours post-dose-NCS;n=0,6,0,0,2 |  | 0 |  |  | 0
  Day 6: 0.5 to 4 hours post-dose-CS;n=0,0,6,0,2: number analyzed (Participants) | 0 | 0 | 6 | 0 | 2
  Day 6: 0.5 to 4 hours post-dose-CS;n=0,0,6,0,2 |  |  | 0 |  | 0
  Day 6: 0.5 to 4 hours post-dose-NCS;n=0,0,6,0,2: number analyzed (Participants) | 0 | 0 | 6 | 0 | 2
  Day 6: 0.5 to 4 hours post-dose-NCS;n=0,0,6,0,2 |  |  | 0 |  | 0
  Day 7: 0.5 to 4 hours post-dose-CS;n=0,0,0,12,2: number analyzed (Participants) | 0 | 0 | 0 | 12 | 2
  Day 7: 0.5 to 4 hours post-dose-CS;n=0,0,0,12,2 |  |  |  | 0 | 0
  Day 7: 0.5 to 4 hours post-dose-NCS;n=0,0,0,12,2: number analyzed (Participants) | 0 | 0 | 0 | 12 | 2
  Day 7: 0.5 to 4 hours post-dose-NCS;n=0,0,0,12,2 |  |  |  | 0 | 0
  Day 12: 0.5 to 4 hours post-dose-CS;n=0,0,6,12,4: number analyzed (Participants) | 0 | 0 | 6 | 12 | 4
  Day 12: 0.5 to 4 hours post-dose-CS;n=0,0,6,12,4 |  |  | 0 | 0 | 0
  Day 12: 0.5 to 4 hours post-dose-NCS;n=0,0,6,12,4: number analyzed (Participants) | 0 | 0 | 6 | 12 | 4
  Day 12: 0.5 to 4 hours post-dose-NCS;n=0,0,6,12,4 |  |  | 0 | 0 | 1
  Day 18: 0.5 to 4 hours post-dose-CS;n=0,0,6,0,2: number analyzed (Participants) | 0 | 0 | 6 | 0 | 2
  Day 18: 0.5 to 4 hours post-dose-CS;n=0,0,6,0,2 |  |  | 0 |  | 0
  Day 18: 0.5 to 4 hours post-dose-NCS;n=0,0,6,0,2: number analyzed (Participants) | 0 | 0 | 6 | 0 | 2
  Day 18: 0.5 to 4 hours post-dose-NCS;n=0,0,6,0,2 |  |  | 0 |  | 0

32. Primary Outcome: Part 2: Number of Participants With Abnormal Telemetry Findings
Description: Continuous cardiac telemetry was performed from approximately 0.5 hour (pre-dose) to 4 hours post-dose. Abnormal findings were categorized as CS and NCS. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: Days 1, 7, 12 and 13: 0.5 hour (pre-dose) to 4 hours post-dose
Population: Safety Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Cohort A- CCI15106 60 mg SD | Part 2: Cohort A- Placebo | Part 2: Cohort B- CCI15106 60 mg BID
Number analyzed (Participants) | 6 | 2 | 8
Participants
  Day 1: 0.5 to 4 hours post-dose-CS; n=6,2,8 | 0 | 0 | 0
  Day 1: 0.5 to 4 hours post-dose-NCS; n=6,2,8 | 0 | 0 | 1
  Day 7: 0.5 to 4 hours post-dose-CS; n=0,0,8: number analyzed (Participants) | 0 | 0 | 8
  Day 7: 0.5 to 4 hours post-dose-CS; n=0,0,8 |  |  | 0
  Day 7: 0.5 to 4 hours post-dose-NCS; n=0,0,8: number analyzed (Participants) | 0 | 0 | 8
  Day 7: 0.5 to 4 hours post-dose-NCS; n=0,0,8 |  |  | 2
  Day 12: 0.5 to 4 hours post-dose-CS; n=0,0,5: number analyzed (Participants) | 0 | 0 | 5
  Day 12: 0.5 to 4 hours post-dose-CS; n=0,0,5 |  |  | 0
  Day 12: 0.5 to 4 hours post-dose-NCS; n=0,0,5: number analyzed (Participants) | 0 | 0 | 5
  Day 12: 0.5 to 4 hours post-dose-NCS; n=0,0,5 |  |  | 0
  Day 13: 0.5 to 4 hours post-dose-CS; n=0,0,3: number analyzed (Participants) | 0 | 0 | 3
  Day 13: 0.5 to 4 hours post-dose-CS; n=0,0,3 |  |  | 0
  Day 13: 0.5 to 4 hours post-dose-NCS; n=0,0,3: number analyzed (Participants) | 0 | 0 | 3
  Day 13: 0.5 to 4 hours post-dose-NCS; n=0,0,3 |  |  | 1

33. Primary Outcome: Part 1: Percent Predicted Forced Expiratory Volume in 1 Second (FEV1) at Indicated Time Points
Description: FEV1 is a measure of lung function and the maximal amount of air that can be forcefully exhaled in one second. FEV1 was measured using standard spirometry. Percent predicted FEV1 was calculated as: Percent predicted FEV1=(maximum FEV1 divided by predicted normal FEV1)*100.
Time Frame: Days 1, 3, 6 and 19: pre-dose, 0.25, 0.5, 1 and 4 hours post-dose; Days 8, 11 and 16: pre-dose and 4 hours post-dose; Day 14: pre-dose, 0.5, 1 and 4 hours post-dose
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Percent predicted FEV1
Arm/Group | Part 1: Cohort A- CCI15106 60 mg SD | Part 1: Cohort A- CCI15106 120 mg SD | Part 1: Cohort A- CCI15106 30 mg BID | Part 1: Cohort B- CCI15106 60 mg BID | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 12 | 4
Percent predicted FEV1
  Day 1: pre-dose, n=6,0,0,12,4: number analyzed (Participants) | 6 | 0 | 0 | 12 | 4
  Day 1: pre-dose, n=6,0,0,12,4 | 101.0 (8.49) |  |  | 101.1 (15.31) | 102.0 (9.35)
  Day 1: 0.25 hour, n=6,0,0,0,2: number analyzed (Participants) | 6 | 0 | 0 | 0 | 2
  Day 1: 0.25 hour, n=6,0,0,0,2 | 101.5 (7.87) |  |  |  | 99.0 (14.14)
  Day 1: 0.5 hour, n=6,0,0,12,4: number analyzed (Participants) | 6 | 0 | 0 | 12 | 4
  Day 1: 0.5 hour, n=6,0,0,12,4 | 104.3 (7.17) |  |  | 100.3 (13.94) | 102.5 (12.82)
  Day 1: 1 hour, n=6,0,0,12,4: number analyzed (Participants) | 6 | 0 | 0 | 12 | 4
  Day 1: 1 hour, n=6,0,0,12,4 | 105.2 (6.62) |  |  | 102.2 (14.86) | 103.8 (11.56)
  Day 1: 4 hours, n=6,0,0,12,4: number analyzed (Participants) | 6 | 0 | 0 | 12 | 4
  Day 1: 4 hours, n=6,0,0,12,4 | 104.5 (8.04) |  |  | 101.4 (16.20) | 104.3 (11.76)
  Day 3: pre-dose, n=0,6,0,12,4: number analyzed (Participants) | 0 | 6 | 0 | 12 | 4
  Day 3: pre-dose, n=0,6,0,12,4 |  | 103.2 (5.71) |  | 101.5 (14.47) | 105.3 (12.45)
  Day 3: 0.25 hour, n=0,6,0,0,2: number analyzed (Participants) | 0 | 6 | 0 | 0 | 2
  Day 3: 0.25 hour, n=0,6,0,0,2 |  | 103.2 (6.49) |  |  | 102.5 (19.09)
  Day 3: 0.5 hour, n=0,6,0,0,2: number analyzed (Participants) | 0 | 6 | 0 | 0 | 2
  Day 3: 0.5 hour, n=0,6,0,0,2 |  | 103.0 (5.97) |  |  | 100.0 (18.38)
  Day 3: 1 hour, n=0,6,0,0,2: number analyzed (Participants) | 0 | 6 | 0 | 0 | 2
  Day 3: 1 hour, n=0,6,0,0,2 |  | 104.3 (6.68) |  |  | 101.0 (16.97)
  Day 3: 4 hours, n=0,6,0,12,4: number analyzed (Participants) | 0 | 6 | 0 | 12 | 4
  Day 3: 4 hours, n=0,6,0,12,4 |  | 106.7 (7.00) |  | 103.1 (15.64) | 106.8 (12.95)
  Day 6: pre-dose, n=0,0,6,12,4: number analyzed (Participants) | 0 | 0 | 6 | 12 | 4
  Day 6: pre-dose, n=0,0,6,12,4 |  |  | 104.5 (5.61) | 101.3 (15.69) | 102.8 (10.94)
  Day 6: 0.25 hour, n=0,0,6,0,2: number analyzed (Participants) | 0 | 0 | 6 | 0 | 2
  Day 6: 0.25 hour, n=0,0,6,0,2 |  |  | 102.3 (6.80) |  | 101.5 (17.68)
  Day 6: 0.5 hour, n=0,0,6,0,2: number analyzed (Participants) | 0 | 0 | 6 | 0 | 2
  Day 6: 0.5 hour, n=0,0,6,0,2 |  |  | 103.5 (7.31) |  | 101.0 (18.38)
  Day 6: 1 hour, n=0,0,6,0,2: number analyzed (Participants) | 0 | 0 | 6 | 0 | 2
  Day 6: 1 hour, n=0,0,6,0,2 |  |  | 104.0 (6.26) |  | 99.0 (18.38)
  Day 6: 4 hours, n=0,0,6,12,4: number analyzed (Participants) | 0 | 0 | 6 | 12 | 4
  Day 6: 4 hours, n=0,0,6,12,4 |  |  | 106.3 (3.93) | 104.0 (15.50) | 105.5 (10.66)
  Day 8: pre-dose, n=0,0,6,0,2: number analyzed (Participants) | 0 | 0 | 6 | 0 | 2
  Day 8: pre-dose, n=0,0,6,0,2 |  |  | 105.0 (5.73) |  | 103.0 (16.97)
  Day 8: 4 hours, n=0,0,6,0,2: number analyzed (Participants) | 0 | 0 | 6 | 0 | 2
  Day 8: 4 hours, n=0,0,6,0,2 |  |  | 104.7 (4.50) |  | 103.5 (17.68)
  Day 11: pre-dose, n=0,0,6,12,4: number analyzed (Participants) | 0 | 0 | 6 | 12 | 4
  Day 11: pre-dose, n=0,0,6,12,4 |  |  | 103.3 (3.88) | 101.6 (16.76) | 106.0 (11.28)
  Day 11: 4 hours, n=0,0,6,12,4: number analyzed (Participants) | 0 | 0 | 6 | 12 | 4
  Day 11: 4 hours, n=0,0,6,12,4 |  |  | 105.0 (6.69) | 103.6 (15.84) | 107.0 (10.42)
  Day 14: pre-dose, n=0,0,0,11,2: number analyzed (Participants) | 0 | 0 | 0 | 11 | 2
  Day 14: pre-dose, n=0,0,0,11,2 |  |  |  | 101.0 (16.84) | 105.5 (6.36)
  Day 14: 0.5 hour, n=0,0,0,11,2: number analyzed (Participants) | 0 | 0 | 0 | 11 | 2
  Day 14: 0.5 hour, n=0,0,0,11,2 |  |  |  | 100.7 (15.88) | 104.0 (8.49)
  Day 14: 1 hour, n=0,0,0,12,2: number analyzed (Participants) | 0 | 0 | 0 | 12 | 2
  Day 14: 1 hour, n=0,0,0,12,2 |  |  |  | 99.1 (16.09) | 107.5 (6.36)
  Day 14: 4 hours, n=0,0,0,12,2: number analyzed (Participants) | 0 | 0 | 0 | 12 | 2
  Day 14: 4 hours, n=0,0,0,12,2 |  |  |  | 97.3 (16.23) | 112.5 (9.19)
  Day 16: pre-dose, n=0,0,6,0,2: number analyzed (Participants) | 0 | 0 | 6 | 0 | 2
  Day 16: pre-dose, n=0,0,6,0,2 |  |  | 102.5 (5.32) |  | 104.5 (17.68)
  Day 16: 4 hours, n=0,0,6,0,2: number analyzed (Participants) | 0 | 0 | 6 | 0 | 2
  Day 16: 4 hours, n=0,0,6,0,2 |  |  | 105.3 (6.38) |  | 104.0 (19.80)
  Day 19: pre-dose, n=0,0,6,0,2: number analyzed (Participants) | 0 | 0 | 6 | 0 | 2
  Day 19: pre-dose, n=0,0,6,0,2 |  |  | 101.7 (7.47) |  | 104.0 (18.38)
  Day 19: 0.25 hour, n=0,0,6,0,2: number analyzed (Participants) | 0 | 0 | 6 | 0 | 2
  Day 19: 0.25 hour, n=0,0,6,0,2 |  |  | 102.5 (6.72) |  | 99.5 (20.51)
  Day 19: 0.5 hour, n=0,0,6,0,2: number analyzed (Participants) | 0 | 0 | 6 | 0 | 2
  Day 19: 0.5 hour, n=0,0,6,0,2 |  |  | 102.7 (10.09) |  | 103.0 (18.38)
  Day 19: 1 hour, n=0,0,6,0,2: number analyzed (Participants) | 0 | 0 | 6 | 0 | 2
  Day 19: 1 hour, n=0,0,6,0,2 |  |  | 99.3 (9.29) |  | 103.5 (16.26)
  Day 19: 4 hours, n=0,0,6,0,2: number analyzed (Participants) | 0 | 0 | 6 | 0 | 2
  Day 19: 4 hours, n=0,0,6,0,2 |  |  | 104.0 (6.78) |  | 103.0 (15.56)

34. Primary Outcome: Part 1: Percent Predicted Forced Vital Capacity (FVC) at Indicated Time Points
Description: FVC is a measure of lung function and the maximal amount of air that can be forcefully exhaled in one second. FVC was measured using standard spirometry. Percent predicted FVC was calculated as: Percent predicted FVC=(maximum FVC divided by predicted normal FVC)*100.
Time Frame: as for outcome 33
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Percent predicted FVC
Arm/Group | Part 1: Cohort A- CCI15106 60 mg SD | Part 1: Cohort A- CCI15106 120 mg SD | Part 1: Cohort A- CCI15106 30 mg BID | Part 1: Cohort B- CCI15106 60 mg BID | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 12 | 4
Percent predicted FVC
  Day 1: pre-dose, n=6,0,0,12,4: number analyzed (Participants) | 6 | 0 | 0 | 12 | 4
  Day 1: pre-dose, n=6,0,0,12,4 | 101.2 (7.14) |  |  | 104.1 (14.19) | 102.0 (2.58)
  Day 1: 0.25 hour, n=6,0,0,0,2: number analyzed (Participants) | 6 | 0 | 0 | 0 | 2
  Day 1: 0.25 hour, n=6,0,0,0,2 | 101.5 (8.41) |  |  |  | 102.0 (5.66)
  Day 1: 0.5 hour, n=6,0,0,12,4: number analyzed (Participants) | 6 | 0 | 0 | 12 | 4
  Day 1: 0.5 hour, n=6,0,0,12,4 | 108.3 (7.31) |  |  | 102.4 (13.28) | 103.8 (2.87)
  Day 1: 1 hour, n=6,0,0,12,4: number analyzed (Participants) | 6 | 0 | 0 | 12 | 4
  Day 1: 1 hour, n=6,0,0,12,4 | 109.8 (7.96) |  |  | 103.7 (13.66) | 105.3 (2.50)
  Day 1: 4 hours, n=6,0,0,12,4: number analyzed (Participants) | 6 | 0 | 0 | 12 | 4
  Day 1: 4 hours, n=6,0,0,12,4 | 106.7 (8.94) |  |  | 103.4 (14.74) | 104.5 (4.36)
  Day 3: pre-dose, n=0,6,0,12,4: number analyzed (Participants) | 0 | 6 | 0 | 12 | 4
  Day 3: pre-dose, n=0,6,0,12,4 |  | 104.3 (6.92) |  | 105.0 (14.68) | 105.8 (2.63)
  Day 3: 0.25 hour, n=0,6,0,0,2: number analyzed (Participants) | 0 | 6 | 0 | 0 | 2
  Day 3: 0.25 hour, n=0,6,0,0,2 |  | 105.7 (8.50) |  |  | 106.5 (3.54)
  Day 3: 0.5 hour, n=0,6,0,0,2: number analyzed (Participants) | 0 | 6 | 0 | 0 | 2
  Day 3: 0.5 hour, n=0,6,0,0,2 |  | 105.0 (8.00) |  |  | 104.5 (3.54)
  Day 3: 1 hour, n=0,6,0,0,2: number analyzed (Participants) | 0 | 6 | 0 | 0 | 2
  Day 3: 1 hour, n=0,6,0,0,2 |  | 105.8 (8.01) |  |  | 105.0 (1.41)
  Day 3: 4 hours, n=0,6,0,12,4: number analyzed (Participants) | 0 | 6 | 0 | 12 | 4
  Day 3: 4 hours, n=0,6,0,12,4 |  | 106.5 (6.72) |  | 105.3 (14.91) | 105.0 (2.16)
  Day 6: pre-dose, n=0,0,6,12,4: number analyzed (Participants) | 0 | 0 | 6 | 12 | 4
  Day 6: pre-dose, n=0,0,6,12,4 |  |  | 107.8 (7.08) | 103.7 (14.77) | 103.3 (2.22)
  Day 6: 0.25 hour, n=0,0,6,0,2: number analyzed (Participants) | 0 | 0 | 6 | 0 | 2
  Day 6: 0.25 hour, n=0,0,6,0,2 |  |  | 104.7 (8.33) |  | 104.5 (2.12)
  Day 6: 0.5 hour, n=0,0,6,0,2: number analyzed (Participants) | 0 | 0 | 6 | 0 | 2
  Day 6: 0.5 hour, n=0,0,6,0,2 |  |  | 105.7 (9.81) |  | 103.5 (2.12)
  Day 6: 1 hour, n=0,0,6,0,2: number analyzed (Participants) | 0 | 0 | 6 | 0 | 2
  Day 6: 1 hour, n=0,0,6,0,2 |  |  | 106.0 (9.14) |  | 99.5 (10.61)
  Day 6: 4 hours, n=0,0,6,12,4: number analyzed (Participants) | 0 | 0 | 6 | 12 | 4
  Day 6: 4 hours, n=0,0,6,12,4 |  |  | 110.2 (7.08) | 105.4 (14.85) | 104.8 (3.30)
  Day 8: pre-dose, n=0,0,6,0,2: number analyzed (Participants) | 0 | 0 | 6 | 0 | 2
  Day 8: pre-dose, n=0,0,6,0,2 |  |  | 108.8 (8.47) |  | 108.0 (1.41)
  Day 8: 4 hours, n=0,0,6,0,2: number analyzed (Participants) | 0 | 0 | 6 | 0 | 2
  Day 8: 4 hours, n=0,0,6,0,2 |  |  | 108.2 (8.47) |  | 108.0 (2.83)
  Day 11: pre-dose, n=0,0,6,12,4: number analyzed (Participants) | 0 | 0 | 6 | 12 | 4
  Day 11: pre-dose, n=0,0,6,12,4 |  |  | 107.2 (7.41) | 104.3 (17.05) | 106.8 (6.13)
  Day 11: 4 hours, n=0,0,6,12,4: number analyzed (Participants) | 0 | 0 | 6 | 12 | 4
  Day 11: 4 hours, n=0,0,6,12,4 |  |  | 107.8 (8.86) | 106.3 (17.43) | 107.0 (5.35)
  Day 14: pre-dose, n=0,0,0,11,2: number analyzed (Participants) | 0 | 0 | 0 | 11 | 2
  Day 14: pre-dose, n=0,0,0,11,2 |  |  |  | 104.7 (16.01) | 102.5 (3.54)
  Day 14: 0.5 hour, n=0,0,0,11,2: number analyzed (Participants) | 0 | 0 | 0 | 11 | 2
  Day 14: 0.5 hour, n=0,0,0,11,2 |  |  |  | 103.6 (14.52) | 100.5 (0.71)
  Day 14: 1 hour, n=0,0,0,12,2: number analyzed (Participants) | 0 | 0 | 0 | 12 | 2
  Day 14: 1 hour, n=0,0,0,12,2 |  |  |  | 100.8 (14.91) | 104.0 (1.41)
  Day 14: 4 hours, n=0,0,0,11,2: number analyzed (Participants) | 0 | 0 | 0 | 11 | 2
  Day 14: 4 hours, n=0,0,0,11,2 |  |  |  | 99.0 (16.81) | 106.0 (0.00)
  Day 16: pre-dose, n=0,0,6,0,2: number analyzed (Participants) | 0 | 0 | 6 | 0 | 2
  Day 16: pre-dose, n=0,0,6,0,2 |  |  | 107.7 (8.04) |  | 111.0 (4.24)
  Day 16: 4 hours, n=0,0,6,0,2: number analyzed (Participants) | 0 | 0 | 6 | 0 | 2
  Day 16: 4 hours, n=0,0,6,0,2 |  |  | 108.5 (8.38) |  | 110.5 (6.36)
  Day 19: pre-dose, n=0,0,6,0,2: number analyzed (Participants) | 0 | 0 | 6 | 0 | 2
  Day 19: pre-dose, n=0,0,6,0,2 |  |  | 104.0 (10.32) |  | 110.0 (4.24)
  Day 19: 0.25 hour, n=0,0,6,0,2: number analyzed (Participants) | 0 | 0 | 6 | 0 | 2
  Day 19: 0.25 hour, n=0,0,6,0,2 |  |  | 105.7 (10.07) |  | 107.0 (7.07)
  Day 19: 0.5 hour, n=0,0,6,0,2: number analyzed (Participants) | 0 | 0 | 6 | 0 | 2
  Day 19: 0.5 hour, n=0,0,6,0,2 |  |  | 104.3 (10.73) |  | 106.5 (7.78)
  Day 19: 1 hour, n=0,0,6,0,2: number analyzed (Participants) | 0 | 0 | 6 | 0 | 2
  Day 19: 1 hour, n=0,0,6,0,2 |  |  | 100.8 (11.84) |  | 103.5 (6.36)
  Day 19: 4 hours, n=0,0,6,0,2: number analyzed (Participants) | 0 | 0 | 6 | 0 | 2
  Day 19: 4 hours, n=0,0,6,0,2 |  |  | 101.0 (8.88) |  | 101.5 (6.36)

35. Primary Outcome: Part 2: Percent Predicted FEV1 at Indicated Time Points
Description: as for outcome 33
Time Frame: Day 1 and 14: pre-dose, 0.25, 0.5, 1 and 4 hours post-dose; Days 3, 6 and 11: pre-dose and 4 hours post-dose
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Percent predicted FEV1
Arm/Group | Part 2: Cohort A- CCI15106 60 mg SD | Part 2: Cohort A- Placebo | Part 2: Cohort B- CCI15106 60 mg BID
Number analyzed (Participants) | 6 | 2 | 8
Percent predicted FEV1
  Day 1: pre-dose, n=6,2,8 | 50.3 (13.88) | 51.5 (20.51) | 52.4 (5.95)
  Day 1: 0.25 hour, n=6,2,8 | 45.3 (10.93) | 41.0 (24.04) | 44.8 (4.13)
  Day 1: 0.5 hour, n=6,2,8 | 47.8 (12.45) | 43.0 (24.04) | 47.8 (4.17)
  Day 1: 1 hour, n=6,2,8 | 50.5 (13.88) | 45.0 (21.21) | 50.8 (2.87)
  Day 1: 4 hours, n=6,2,8 | 55.5 (12.05) | 50.5 (17.68) | 59.0 (6.30)
  Day 3: pre-dose, n=0,0,8: number analyzed (Participants) | 0 | 0 | 8
  Day 3: pre-dose, n=0,0,8 |  |  | 54.9 (6.71)
  Day 3: 4 hours, n=0,0,8: number analyzed (Participants) | 0 | 0 | 8
  Day 3: 4 hours, n=0,0,8 |  |  | 55.5 (6.44)
  Day 6: pre-dose, n=0,0,8: number analyzed (Participants) | 0 | 0 | 8
  Day 6: pre-dose, n=0,0,8 |  |  | 54.1 (5.28)
  Day 6: 4 hours, n=0,0,8: number analyzed (Participants) | 0 | 0 | 8
  Day 6: 4 hours, n=0,0,8 |  |  | 57.1 (7.57)
  Day 11: pre-dose, n=0,0,8: number analyzed (Participants) | 0 | 0 | 8
  Day 11: pre-dose, n=0,0,8 |  |  | 52.4 (9.65)
  Day 11: 4 hours, n=0,0,8: number analyzed (Participants) | 0 | 0 | 8
  Day 11: 4 hours, n=0,0,8 |  |  | 54.9 (8.54)
  Day 14: pre-dose, n=0,0,8: number analyzed (Participants) | 0 | 0 | 8
  Day 14: pre-dose, n=0,0,8 |  |  | 51.6 (8.31)
  Day 14: 0.25 hour, n=0,0,8: number analyzed (Participants) | 0 | 0 | 8
  Day 14: 0.25 hour, n=0,0,8 |  |  | 46.0 (9.94)
  Day 14: 0.5 hour, n=0,0,8: number analyzed (Participants) | 0 | 0 | 8
  Day 14: 0.5 hour, n=0,0,8 |  |  | 48.1 (8.89)
  Day 14: 1 hour, n=0,0,8: number analyzed (Participants) | 0 | 0 | 8
  Day 14: 1 hour, n=0,0,8 |  |  | 50.3 (8.08)
  Day 14: 4 hours, n=0,0,8: number analyzed (Participants) | 0 | 0 | 8
  Day 14: 4 hours, n=0,0,8 |  |  | 55.6 (6.89)

36. Primary Outcome: Part 2: Percent Predicted FVC at Indicated Time Points
Description: as for outcome 34
Time Frame: Day 1 and 14: pre-dose, 0.25, 0.5, 1 and 4 hours post-dose; Days 3, 6 and 11: pre-dose and 4 hours post-dose
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Percent predicted FVC
Arm/Group | Part 2: Cohort A- CCI15106 60 mg SD | Part 2: Cohort A- Placebo | Part 2: Cohort B- CCI15106 60 mg BID
Number analyzed (Participants) | 6 | 2 | 8
Percent predicted FVC
  Day 1: pre-dose, n=6,2,8 | 74.5 (19.07) | 89.0 (2.83) | 82.8 (15.04)
  Day 1: 0.25 hour, n=6,2,8 | 72.5 (20.03) | 70.5 (10.61) | 76.6 (11.07)
  Day 1: 0.5 hour, n=6,2,8 | 74.7 (18.48) | 76.0 (9.90) | 80.8 (13.49)
  Day 1: 1 hour, n=6,2,8 | 76.7 (20.49) | 77.5 (3.54) | 81.6 (10.14)
  Day 1: 4 hours, n=6,2,8 | 82.0 (15.59) | 91.5 (2.12) | 92.4 (13.31)
  Day 3: pre-dose, n=0,0,8: number analyzed (Participants) | 0 | 0 | 8
  Day 3: pre-dose, n=0,0,8 |  |  | 86.8 (12.33)
  Day 3: 4 hours, n=0,0,8: number analyzed (Participants) | 0 | 0 | 8
  Day 3: 4 hours, n=0,0,8 |  |  | 90.0 (15.01)
  Day 6: pre-dose, n=0,0,8: number analyzed (Participants) | 0 | 0 | 8
  Day 6: pre-dose, n=0,0,8 |  |  | 79.6 (8.72)
  Day 6: 4 hours, n=0,0,8: number analyzed (Participants) | 0 | 0 | 8
  Day 6: 4 hours, n=0,0,8 |  |  | 84.8 (13.26)
  Day 11: pre-dose, n=0,0,8: number analyzed (Participants) | 0 | 0 | 8
  Day 11: pre-dose, n=0,0,8 |  |  | 79.3 (15.78)
  Day 11: 4 hours, n=0,0,8: number analyzed (Participants) | 0 | 0 | 8
  Day 11: 4 hours, n=0,0,8 |  |  | 86.0 (16.67)
  Day 14: pre-dose, n=0,0,8: number analyzed (Participants) | 0 | 0 | 8
  Day 14: pre-dose, n=0,0,8 |  |  | 84.6 (19.59)
  Day 14: 0.25 hour, n=0,0,8: number analyzed (Participants) | 0 | 0 | 8
  Day 14: 0.25 hour, n=0,0,8 |  |  | 76.8 (24.17)
  Day 14: 0.5 hour, n=0,0,8: number analyzed (Participants) | 0 | 0 | 8
  Day 14: 0.5 hour, n=0,0,8 |  |  | 80.3 (24.28)
  Day 14: 1 hour, n=0,0,8: number analyzed (Participants) | 0 | 0 | 8
  Day 14: 1 hour, n=0,0,8 |  |  | 82.9 (25.01)
  Day 14: 4 hours, n=0,0,8: number analyzed (Participants) | 0 | 0 | 8
  Day 14: 4 hours, n=0,0,8 |  |  | 89.1 (17.24)

37. Primary Outcome: Part 1: Number of Participants With Vital Signs Values of PCI
Description: PCI ranges for the vital signs parameters were as follows: systolic blood pressure (SBP) <85 and >160 millimeters of mercury (mmHg), diastolic blood pressure (DBP) <45 and >100 mmHg and heart rate <40 and >110 beats per minute (bpm). Data for the participants with high and low values has been reported.
Time Frame: Up to 51 days
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort A- CCI15106 60 mg SD | Part 1: Cohort A- CCI15106 120 mg SD | Part 1: Cohort A- CCI15106 30 mg BID | Part 1: Cohort B- CCI15106 60 mg BID | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 12 | 4
Participants
  DBP: low | 0 | 0 | 0 | 0 | 0
  DBP: high | 0 | 0 | 0 | 0 | 0
  SBP: low | 0 | 0 | 0 | 0 | 0
  SBP: high | 0 | 0 | 0 | 0 | 0
  Heart rate: low | 0 | 0 | 0 | 0 | 0
  Heart rate: high | 0 | 0 | 0 | 0 | 0

38. Primary Outcome: Part 1: Number of Participants With Vital Signs Values of PCI in Bystanders
Description: PCI ranges for the vital signs parameters were as follows: SBP <85 and >160 mmHg, DBP <45 and >100 mmHg and heart rate <40 and >110 bpm. Data for the participants with high and low values has been reported.
Time Frame: Up to 46 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort C- Bystanders
Number analyzed (Participants) | 14
Participants
  DBP: low | 1
  DBP: high | 0
  SBP: low | 1
  SBP: high | 0
  Heart rate: low | 0
  Heart rate: high | 0

39. Primary Outcome: Part 2: Number of Participants With Vital Signs Values of PCI
Description: as for outcome 38
Time Frame: Up to 46 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Cohort A- CCI15106 60 mg SD | Part 2: Cohort A- Placebo | Part 2: Cohort B- CCI15106 60 mg BID
Number analyzed (Participants) | 6 | 2 | 8
Participants
  DBP: low | 0 | 0 | 0
  DBP: high | 0 | 0 | 0
  SBP: low | 0 | 0 | 0
  SBP: high | 0 | 0 | 1
  Heart rate: low | 0 | 0 | 0
  Heart rate: high | 0 | 0 | 0

40. Primary Outcome: Part 1 Cohort A: Area Under the Curve (AUC) From Time Zero to the Time of Last Quantifiable Concentration (AUC[0-t]) After Single Dose Administration of CCI15106 60 mg on Day 1
Description: Blood samples were collected to evaluate the pharmacokinetics (PKs) of CCI15106 at the indicated time points on Day 1 for the analysis of AUC(0-t) data. PK population consisted of participants who received at least one dose of study treatment and who undergo plasma PK sampling and had at least one post-dose concentration result.
Time Frame: Day 1: pre-dose, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 10, 12, 24 and 48 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part 1: Cohort A- CCI15106 60 mg SD
Number analyzed (Participants) | 6
Hours*nanogram per milliliter | 1255.3711 (19.4)

41. Primary Outcome: Part 1 Cohort A: AUC(0-t) After Single Dose Administration of CCI15106 120 mg on Day 3
Description: Blood samples were collected to evaluate the PKs of CCI15106 at the indicated time points on Day 3 for the analysis of AUC(0-t) data.
Time Frame: Day 3: pre-dose, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 10, 12, 24, 48 and 72 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part 1: Cohort A- CCI15106 120 mg SD
Number analyzed (Participants) | 6
Hours*nanogram per milliliter | 3256.6746 (29.7)

42. Primary Outcome: Part 2 Cohort A: AUC(0-t) After Single Dose Administration of CCI15106 60 mg on Day 1
Description: Blood samples were collected to evaluate the PKs of CCI15106 at the indicated time points on Day 1 for the analysis of AUC(0-t) data.
Time Frame: Day 1: pre-dose, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 10, 12 and 24 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part 2: Cohort A- CCI15106 60 mg SD
Number analyzed (Participants) | 6
Hours*nanogram per milliliter | 862.7642 (59.1)

43. Primary Outcome: Part 1 Cohort A: Maximum Observed Plasma Concentration (Cmax) After Single Dose Administration of CCI15106 60 mg on Day 1
Description: Blood samples were collected to evaluate the PKs of CCI15106 at the indicated time points on Day 1 for the analysis of Cmax data.
Time Frame: Day 1: pre-dose, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 10, 12, 24 and 48 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part 1: Cohort A- CCI15106 60 mg SD
Number analyzed (Participants) | 6
Nanogram per milliliter | 232.2 (20.2)

44. Primary Outcome: Part 1 Cohort A: Cmax After Single Dose Administration of CCI15106 120 mg on Day 3
Description: Blood samples were collected to evaluate the PKs of CCI15106 at the indicated time points on Day 3 for the analysis of Cmax data.
Time Frame: Day 3: pre-dose, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 10, 12, 24, 48 and 72 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part 1: Cohort A- CCI15106 120 mg SD
Number analyzed (Participants) | 6
Nanogram per milliliter | 507.6 (27.6)

45. Primary Outcome: Part 2 Cohort A: Cmax After Single Dose Administration of CCI15106 60 mg on Day 1
Description: as for outcome 43
Time Frame: Day 1: pre-dose, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 10, 12 and 24 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part 2: Cohort A- CCI15106 60 mg SD
Number analyzed (Participants) | 6
Nanogram per milliliter | 179.3 (81.3)

46. Primary Outcome: Part 1 Cohort A: Time of Maximum Concentration (Tmax) After Single Dose Administration of CCI15106 60 mg on Day 1
Description: Blood samples were collected to evaluate the PKs of CCI15106 at the indicated time points on Day 1 for the analysis of tmax data.
Time Frame: Day 1: pre-dose, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 10, 12, 24 and 48 hours post-dose
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: Cohort A- CCI15106 60 mg SD
Number analyzed (Participants) | 6
Hours | 0.500 [0.25 to 1.00]

47. Primary Outcome: Part 1 Cohort A: Tmax After Single Dose Administration of CCI15106 120 mg on Day 3
Description: Blood samples were collected to evaluate the PKs of CCI15106 at the indicated time points on Day 3 for the analysis of tmax data.
Time Frame: Day 3: pre-dose, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 10, 12, 24, 48 and 72 hours post-dose
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: Cohort A- CCI15106 120 mg SD
Number analyzed (Participants) | 6
Hours | 0.625 [0.25 to 0.75]

48. Primary Outcome: Part 2 Cohort A: Tmax After Single Dose Administration of CCI15106 60 mg on Day 1
Description: as for outcome 46
Time Frame: Day 1: pre-dose, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 10, 12 and 24 hours post-dose
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2: Cohort A- CCI15106 60 mg SD
Number analyzed (Participants) | 6
Hours | 0.500 [0.27 to 0.75]

49. Primary Outcome: Part 1 Cohort A: AUC From Time Zero to Infinity (AUC[0-infinity]) After Single Dose Administration of CCI15106 60 mg on Day 1
Description: Blood samples were collected to evaluate the PKs of CCI15106 at the indicated time points on Day 1 for the analysis of AUC(0-infinity) data.
Time Frame: Day 1: pre-dose, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 10, 12, 24 and 48 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part 1: Cohort A- CCI15106 60 mg SD
Number analyzed (Participants) | 6
Hours*nanogram per milliliter | 1618.4216 (20.6)

50. Primary Outcome: Part 1 Cohort A: AUC(0-infinity) After Single Dose Administration of CCI15106 120 mg on Day 3
Description: Blood samples were collected to evaluate the PKs of CCI15106 at the indicated time points on Day 3 for the analysis of AUC(0-infinity) data.
Time Frame: Day 3: pre-dose, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 10, 12, 24, 48 and 72 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part 1: Cohort A- CCI15106 120 mg SD
Number analyzed (Participants) | 6
Hours*nanogram per milliliter | 4418.9437 (37.7)

51. Primary Outcome: Part 2 Cohort A: AUC(0-infinity) After Single Dose Administration of CCI15106 60 mg on Day 1
Description: as for outcome 49
Time Frame: Day 1: pre-dose, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 10, 12 and 24 hours post-dose
Population: PK Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part 2: Cohort A- CCI15106 60 mg SD
Number analyzed (Participants) | 4
Hours*nanogram per milliliter | 968.8838 (49.4)

52. Primary Outcome: Part 1 Cohort A: Elimination Half-life (t1/2) After Single Dose Administration of CCI15106 60 mg on Day 1
Description: Blood samples were collected to evaluate the PKs of CCI15106 at the indicated time points on Day 1 for the analysis of t1/2 data.
Time Frame: Day 1: pre-dose, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 10, 12, 24 and 48 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1: Cohort A- CCI15106 60 mg SD
Number analyzed (Participants) | 6
Hours | 25.8346 (5.1)

53. Primary Outcome: Part 1 Cohort A: t1/2 After Single Dose Administration of CCI15106 120 mg on Day 3
Description: Blood samples were collected to evaluate the PKs of CCI15106 at the indicated time points on Day 3 for the analysis of t1/2 data.
Time Frame: Day 3: pre-dose, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 10, 12, 24, 48 and 72 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1: Cohort A- CCI15106 120 mg SD
Number analyzed (Participants) | 6
Hours | 41.2596 (32.0)

54. Primary Outcome: Part 2 Cohort A: t1/2 After Single Dose Administration of CCI15106 60 mg on Day 1
Description: as for outcome 52
Time Frame: Day 1: pre-dose, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 10, 12 and 24 hours post-dose
Population: PK Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 2: Cohort A- CCI15106 60 mg SD
Number analyzed (Participants) | 4
Hours | 16.4000 (8.3)

55. Primary Outcome: Part 1 Cohort A: Clearance (CL/F) After Single Dose Administration of CCI15106 60 mg on Day 1
Description: Blood samples were collected to evaluate the PKs of CCI15106 at the indicated time points on Day 1 for the analysis of CL/F data.
Time Frame: Day 1: pre-dose, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 10, 12, 24 and 48 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Part 1: Cohort A- CCI15106 60 mg SD
Number analyzed (Participants) | 6
Liters per hour | 37.0732 (20.6)

56. Primary Outcome: Part 1 Cohort A: CL/F After Single Dose Administration of CCI15106 120 mg on Day 3
Description: Blood samples were collected to evaluate the PKs of CCI15106 at the indicated time points on Day 3 for the analysis of CL/F data.
Time Frame: Day 3: pre-dose, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 10, 12, 24, 48 and 72 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Part 1: Cohort A- CCI15106 120 mg SD
Number analyzed (Participants) | 6
Liters per hour | 27.1558 (37.7)

57. Primary Outcome: Part 2 Cohort A: CL/F After Single Dose Administration of CCI15106 60 mg on Day 1
Description: as for outcome 55
Time Frame: Day 1: pre-dose, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 10, 12 and 24 hours post-dose
Population: PK Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Part 2: Cohort A- CCI15106 60 mg SD
Number analyzed (Participants) | 4
Liters per hour | 61.9269 (49.4)

58. Primary Outcome: Part 1 Cohort A: AUC From Time Zero to End of Dosing Interval (AUC[0-tau]) After Repeated Dose Administration of CCI15106 30 mg
Description: Blood samples were collected to evaluate the PKs of CCI15106 at the indicated time points on Days 6 and 19 for the analysis of AUC(0-tau) data.
Time Frame: Day 6: pre-dose, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 10 and 12 hours post-dose; Day 19: pre-dose, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 10, 12, 24, 48 and 72 hours post-dose
Population: PK Population. NA indicates that, AUC(0-tau) could not be calculated because t1/2 considered unreliable as period over which they were calculated was less than twice resultant t1/2 in all cases. In addition, percent AUCextrapolated (%AUCex) was >20% in most cases. This was largely due to short period of sampling times.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part 1: Cohort A- CCI15106 30 mg BID
Number analyzed (Participants) | 6
Hours*nanogram per milliliter
  Day 6 | NA (NA) — AUC(0-tau) could not be calculated because t1/2 considered unreliable as period over which they were calculated was < twice resultant t1/2 in all cases.In addition,%AUCex was >20% in most cases.This was largely due to short period of sampling times.
  Day 19 | 1214.2671 (21.1)

59. Primary Outcome: Part 1 Cohort B: AUC(0-tau) After Repeated Dose Administration of CCI15106 60 mg
Description: Blood samples were collected to evaluate the PKs of CCI15106 at the indicated time points on Days 1 and 14 for the analysis of AUC(0-tau) data.
Time Frame: Days 1 and 14: pre-dose, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 10 and 12 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part 1: Cohort B- CCI15106 60 mg BID
Number analyzed (Participants) | 12
Hours*nanogram per milliliter
  Day 1, n=12 | 564.7314 (50.2)
  Day 14, n=8: number analyzed (Participants) | 8
  Day 14, n=8 | 2059.8983 (15.2)

60. Primary Outcome: Part 2 Cohort B: AUC(0-tau) After Repeated Dose Administration of CCI15106 60 mg
Description: as for outcome 59
Time Frame: Days 1 and 14: pre-dose, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 10 and 12 hours post-dose
Population: as for outcome 59
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part 2: Cohort B- CCI15106 60 mg BID
Number analyzed (Participants) | 8
Hours*nanogram per milliliter
  Day 1, n=8 | 687.0875 (39.8)
  Day 14, n=7: number analyzed (Participants) | 7
  Day 14, n=7 | 3086.5172 (28.1)

61. Primary Outcome: Part 1 Cohort A: Cmax After Repeated Dose Administration of CCI15106 30 mg
Description: Blood samples were collected to evaluate the PKs of CCI15106 at the indicated time points on Days 6 and 19 for the analysis of Cmax data.
Time Frame: as for outcome 58
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part 1: Cohort A- CCI15106 30 mg BID
Number analyzed (Participants) | 6
Nanogram per milliliter
  Day 6 | 143.1 (23.2)
  Day 19 | 193.9 (15.1)

62. Primary Outcome: Part 1 Cohort B: Cmax After Repeated Dose Administration of CCI15106 60 mg
Description: Blood samples were collected to evaluate the PKs of CCI15106 at the indicated time points on Days 1 and 14 for the analysis of Cmax data.
Time Frame: Day 1: pre-dose, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 10 and 12 hours post-dose; Day 14: pre-dose, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 10, 12 and 24 hours post-dose
Population: as for outcome 59
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part 1: Cohort B- CCI15106 60 mg BID
Number analyzed (Participants) | 12
Nanogram per milliliter
  Day 1, n=12 | 188.7 (63.5)
  Day 14, n=11: number analyzed (Participants) | 11
  Day 14, n=11 | 285.0 (39.0)

63. Primary Outcome: Part 2 Cohort B: Cmax After Repeated Dose Administration of CCI15106 60 mg
Description: as for outcome 62
Time Frame: Day 1: pre-dose, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 10 and 12 hours post-dose; Day14: pre-dose, 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 10, 12 and 24 hours post-dose
Population: PK Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part 2: Cohort B- CCI15106 60 mg BID
Number analyzed (Participants) | 8
Nanogram per milliliter
  Day 1 | 178.2 (51.4)
  Day 14 | 423.0 (31.9)

64. Primary Outcome: Part 1 Cohort A: Tmax After Repeated Dose Administration of CCI15106 30 mg
Description: Blood samples were collected to evaluate the PKs of CCI15106 at the indicated time points on Days 6 and 19 for the analysis of tmax data.
Time Frame: as for outcome 58
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: Cohort A- CCI15106 30 mg BID
Number analyzed (Participants) | 6
Hours
  Day 6 | 0.500 [0.50 to 0.75]
  Day 19 | 0.500 [0.25 to 0.50]

65. Primary Outcome: Part 1 Cohort B: Tmax After Repeated Dose Administration of CCI15106 60 mg
Description: Blood samples were collected to evaluate the PKs of CCI15106 at the indicated time points on Days 1 and 14 for the analysis of tmax data.
Time Frame: as for outcome 62
Population: as for outcome 59
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: Cohort B- CCI15106 60 mg BID
Number analyzed (Participants) | 12
Hours
  Day 1, n=12 | 0.633 [0.50 to 1.00]
  Day 14, n=11: number analyzed (Participants) | 11
  Day 14, n=11 | 0.500 [0.30 to 1.00]

66. Primary Outcome: Part 2 Cohort B: Tmax After Repeated Dose Administration of CCI15106 60 mg
Description: as for outcome 65
Time Frame: as for outcome 63
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2: Cohort B- CCI15106 60 mg BID
Number analyzed (Participants) | 8
Hours
  Day 1 | 0.633 [0.25 to 1.00]
  Day 14 | 0.500 [0.25 to 1.00]

67. Primary Outcome: Part 1 Cohort A: t1/2 After Repeated Dose Administration of CCI15106 30 mg
Description: Blood samples were collected to evaluate the PKs of CCI15106 at the indicated time points on Days 6 and 19 for the analysis of t1/2 data.
Time Frame: as for outcome 58
Population: PK Population. NA indicates that, t1/2 of CCI15106 plasma concentration in healthy participant was estimated but considered unreliable as period over which they were calculated was less than twice resultant t1/2 in all cases. In addition, %AUCex was >20% in most cases. This was largely due to short period of sampling times.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1: Cohort A- CCI15106 30 mg BID
Number analyzed (Participants) | 6
Hours
  Day 6 | NA (NA) — t1/2 of CCI15106 plasma concentration was estimated but considered unreliable as period over which they were calculated was < twice resultant t1/2 in all cases.%AUCex was >20% in most cases.This was largely due to short period of sampling times.
  Day 19 | 18.1484 (10.2)

68. Primary Outcome: Part 1 Cohort B: t1/2 After Repeated Dose Administration of CCI15106 60 mg
Description: Blood samples were collected to evaluate the PKs of CCI15106 at the indicated time points on Days 1 and 14 for the analysis of t1/2 data.
Time Frame: as for outcome 62
Population: as for outcome 59
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1: Cohort B- CCI15106 60 mg BID
Number analyzed (Participants) | 12
Hours
  Day 1, n=12 | 8.3719 (14.2)
  Day 14, n=8: number analyzed (Participants) | 8
  Day 14, n=8 | 23.0497 (42.4)

69. Primary Outcome: Part 2 Cohort B: t1/2 After Repeated Dose Administration of CCI15106 60 mg
Description: as for outcome 68
Time Frame: as for outcome 63
Population: as for outcome 59
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 2: Cohort B- CCI15106 60 mg BID
Number analyzed (Participants) | 8
Hours
  Day 1, n=8 | 8.1572 (18.0)
  Day 14, n=7: number analyzed (Participants) | 7
  Day 14, n=7 | 21.5034 (39.6)

70. Primary Outcome: Part 1: Concentration of CCI15106 in Plasma of Bystanders: Cohort C
Description: Blood samples were collected from bystanders 15 minutes after dosing at indicated time points. Bystander PK population consisted of participants who were present at least once in the room with the participant receiving the dose, undergo plasma PK sampling and had post-dose concentration result.
Time Frame: Days 1, 7 and 14: pre-dose, 15 minutes post-dose
Population: Bystander PK Population. NA indicates that, data could not be analyzed because data was below level of quantification.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | Part 1: Cohort C- Bystanders
Number analyzed (Participants) | 14
Nanogram per milliliter | NA (NA) — Data could not be analyzed because data was below level of quantification.

71. Primary Outcome: Part 1: Concentration of CCI15106 Accumulated on Filters Fitted on Bystander: Cohort C
Description: Personal exposure air samples were collected on filters placed on each bystander after the first daily dose at indicated time points. The filters were used to measure CCI15106 concentration in the person's breathing zone. Fixed location concentrations were measured near window, near door, back to wall and facing wall in the dosing room over 15 minutes post-dose. Each bystander had a filter attached to their study clothing. The filters were measured for CCI15106. This was a single measurement from the filter for each bystsander. The locations (near window, near door, back to wall and facing wall) were just to record where the bystander was located in the room.
Time Frame: Days 1, 7 and 14: 15 minutes post-dose
Population: Bystander PK Population. Only those participants with data available at the specified time points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Microgram per cubic meter
Groups:
- Part 1: Bystander Group 1- Session 1; Part 1: Bystander Group 2- Session 1: Participants inhaled the dose of CCI15106 60 mg BID via Monodose RS01 in a room designated for dosing. Only participants inhaled the dose and designated bystanders (healthy participants enrolled to evaluate bystander exposure) were allowed in the room during inhalation of the airborne drug in session 1 on Days 1, 7 and 14.
- Part 1: Bystander Group 1- Session 2; Part 1: Bystander Group 4- Session 2: Participants inhaled the dose of CCI15106 60 mg BID via Monodose RS01 in a room designated for dosing. Only participants inhaled the dose and designated bystanders (healthy participants enrolled to evaluate bystander exposure) were allowed in the room during inhalation of the airborne drug in session 2 on Days 1, 7 and 14.
- Part 1: Bystander Group 2- Session 2: Participants inhaled the dose of CCI15106 60 mg or matching placebo BID via Monodose RS01 in a room designated for dosing. Only participants inhaled the dose and designated bystanders (healthy participants enrolled to evaluate bystander exposure) were allowed in the room during inhalation of the airborne drug in session 2 on Days 1, 7 and 14.
- Part 1: Bystander Group 3- Session 1: Participants inhaled the dose of CCI15106 60 mg BID via Monodose RS01 in a room designated for dosing. Only participants inhaled the dose and designated bystanders (healthy participants enrolled to evaluate bystander exposure) were allowed in the room during inhalation of the airborne drug in a single session on Days 1, 7 and 14.
- Part 1: Bystander Group 4- Session 1: Participants inhaled the dose of CCI15106 60 mg or matching placebo BID via Monodose RS01 in a room designated for dosing. Only participants inhaled the dose and designated bystanders (healthy participants enrolled to evaluate bystander exposure) were allowed in the room during inhalation of the airborne drug in session 1 on Days 1, 7 and 14.
Arm/Group | Part 1: Bystander Group 1- Session 1 | Part 1: Bystander Group 1- Session 2 | Part 1: Bystander Group 2- Session 1 | Part 1: Bystander Group 2- Session 2 | Part 1: Bystander Group 3- Session 1 | Part 1: Bystander Group 4- Session 1 | Part 1: Bystander Group 4- Session 2
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 2
Microgram per cubic meter
  Day 1: Near door,n=1,1,1,1,0,0,0: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 0 | 0
  Day 1: Near door,n=1,1,1,1,0,0,0 | 0.53 (NA) — Standard deviation could not be calculated for one participant. | 0.39 (NA) — Standard deviation could not be calculated for one participant. | 1.81 (NA) — Standard deviation could not be calculated for one participant. | 8.99 (NA) — Standard deviation could not be calculated for one participant. |  |  |
  Day 1: Near window,n=1,1,1,1,0,0,0: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 0 | 0
  Day 1: Near window,n=1,1,1,1,0,0,0 | 1.10 (NA) — Standard deviation could not be calculated for one participant. | 0.10 (NA) — Standard deviation could not be calculated for one participant. | 2.46 (NA) — Standard deviation could not be calculated for one participant. | 4.84 (NA) — Standard deviation could not be calculated for one participant. |  |  |
  Day 1: Back to wall,n=0,0,0,0,1,1,1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 1
  Day 1: Back to wall,n=0,0,0,0,1,1,1 |  |  |  |  | 5.27 (NA) — Standard deviation could not be calculated for one participant. | 0.10 (NA) — Standard deviation could not be calculated for one participant. | 0.10 (NA) — Standard deviation could not be calculated for one participant.
  Day 1: Facing wall,n=0,0,0,0,1,1,1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 1
  Day 1: Facing wall,n=0,0,0,0,1,1,1 |  |  |  |  | 5.84 (NA) — Standard deviation could not be calculated for one participant. | 0.10 (NA) — Standard deviation could not be calculated for one participant. | 0.10 (NA) — Standard deviation could not be calculated for one participant.
  Day 7: Near door,n=1,1,1,1,0,0,0: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 0 | 0
  Day 7: Near door,n=1,1,1,1,0,0,0 | 2.81 (NA) — Standard deviation could not be calculated for one participant. | 2.62 (NA) — Standard deviation could not be calculated for one participant. | 2.13 (NA) — Standard deviation could not be calculated for one participant. | 0.49 (NA) — Standard deviation could not be calculated for one participant. |  |  |
  Day 7: Near window,n=1,1,1,1,0,0,0: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 0 | 0
  Day 7: Near window,n=1,1,1,1,0,0,0 | 2.86 (NA) — Standard deviation could not be calculated for one participant. | 2.74 (NA) — Standard deviation could not be calculated for one participant. | 3.14 (NA) — Standard deviation could not be calculated for one participant. | 0.41 (NA) — Standard deviation could not be calculated for one participant. |  |  |
  Day 7: Back to wall,n=0,0,0,0,1,1,1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 1
  Day 7: Back to wall,n=0,0,0,0,1,1,1 |  |  |  |  | 0.76 (NA) — Standard deviation could not be calculated for one participant. | 0.47 (NA) — Standard deviation could not be calculated for one participant. | 0.80 (NA) — Standard deviation could not be calculated for one participant.
  Day 7: Facing wall,n=0,0,0,0,1,1,1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 1
  Day 7: Facing wall,n=0,0,0,0,1,1,1 |  |  |  |  | 0.86 (NA) — Standard deviation could not be calculated for one participant. | 0.10 (NA) — Standard deviation could not be calculated for one participant. | 1.00 (NA) — Standard deviation could not be calculated for one participant.
  Day 14: Near door,n=1,1,1,1,0,0,0: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 0 | 0
  Day 14: Near door,n=1,1,1,1,0,0,0 | 0.10 (NA) — Standard deviation could not be calculated for one participant. | 1.97 (NA) — Standard deviation could not be calculated for one participant. | 9.22 (NA) — Standard deviation could not be calculated for one participant. | 0.10 (NA) — Standard deviation could not be calculated for one participant. |  |  |
  Day 14: Near window,n=1,1,1,1,0,0,0: number analyzed (Participants) | 1 | 1 | 1 | 1 | 0 | 0 | 0
  Day 14: Near window,n=1,1,1,1,0,0,0 | 0.10 (NA) — Standard deviation could not be calculated for one participant. | 1.73 (NA) — Standard deviation could not be calculated for one participant. | 8.09 (NA) — Standard deviation could not be calculated for one participant. | 0.45 (NA) — Standard deviation could not be calculated for one participant. |  |  |
  Day 14: Back to wall,n=0,0,0,0,1,1,1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 1
  Day 14: Back to wall,n=0,0,0,0,1,1,1 |  |  |  |  | 0.38 (NA) — Standard deviation could not be calculated for one participant. | 0.35 (NA) — Standard deviation could not be calculated for one participant. | 0.10 (NA) — Standard deviation could not be calculated for one participant.
  Day 14: Facing wall,n=0,0,0,0,1,1,1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 1
  Day 14: Facing wall,n=0,0,0,0,1,1,1 |  |  |  |  | 0.10 (NA) — Standard deviation could not be calculated for one participant. | 0.10 (NA) — Standard deviation could not be calculated for one participant. | 0.10 (NA) — Standard deviation could not be calculated for one participant.

72. Primary Outcome: Part 1: Concentration of CCI15106 Accumulated on Filters Fitted on Stationary Pumps: Cohort C
Description: Static air samples were collected on filters within air pumps positioned in two locations (bench and corner) in the room. Sampling devices attached to sampling pumps were used to measure CCI15106 concentration. Fixed location concentrations were measured in corner of room and on bench at back of room over 20 minutes and 60 minutes post-dosing.
Time Frame: Days 1, 7 and 14: 20 and 60 minutes post-dose
Population: Bystander PK Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Microgram per cubic meter
Arm/Group | Part 1: Bystander Group 1- Session 1 | Part 1: Bystander Group 1- Session 2 | Part 1: Bystander Group 2- Session 1 | Part 1: Bystander Group 2- Session 2 | Part 1: Bystander Group 3- Session 1 | Part 1: Bystander Group 4- Session 1 | Part 1: Bystander Group 4- Session 2
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 2
Microgram per cubic meter
  Day 1: 20 minutes- Corner,n=1,1,1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1
  Day 1: 20 minutes- Corner,n=1,1,1,1,1,1,1 | 0.79 (NA) — Standard deviation could not be calculated for one participant. | 0.50 (NA) — Standard deviation could not be calculated for one participant. | 2.09 (NA) — Standard deviation could not be calculated for one participant. | 4.12 (NA) — Standard deviation could not be calculated for one participant. | 5.80 (NA) — Standard deviation could not be calculated for one participant. | 0.50 (NA) — Standard deviation could not be calculated for one participant. | 0.50 (NA) — Standard deviation could not be calculated for one participant.
  Day 1: 20 minutes- Bench,n=1,1,1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1
  Day 1: 20 minutes- Bench,n=1,1,1,1,1,1,1 | 1.46 (NA) — Standard deviation could not be calculated for one participant. | 0.50 (NA) — Standard deviation could not be calculated for one participant. | 1.58 (NA) — Standard deviation could not be calculated for one participant. | 3.74 (NA) — Standard deviation could not be calculated for one participant. | 4.98 (NA) — Standard deviation could not be calculated for one participant. | 0.50 (NA) — Standard deviation could not be calculated for one participant. | 0.50 (NA) — Standard deviation could not be calculated for one participant.
  Day 7: 20 minutes- Corner,n=1,1,1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1
  Day 7: 20 minutes- Corner,n=1,1,1,1,1,1,1 | 1.52 (NA) — Standard deviation could not be calculated for one participant. | 2.53 (NA) — Standard deviation could not be calculated for one participant. | 2.64 (NA) — Standard deviation could not be calculated for one participant. | 0.30 (NA) — Standard deviation could not be calculated for one participant. | 0.30 (NA) — Standard deviation could not be calculated for one participant. | 0.28 (NA) — Standard deviation could not be calculated for one participant. | 1.01 (NA) — Standard deviation could not be calculated for one participant.
  Day 7: 20 minutes- Bench,n=1,1,1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1
  Day 7: 20 minutes- Bench,n=1,1,1,1,1,1,1 | 2.39 (NA) — Standard deviation could not be calculated for one participant. | 3.32 (NA) — Standard deviation could not be calculated for one participant. | 2.34 (NA) — Standard deviation could not be calculated for one participant. | 0.46 (NA) — Standard deviation could not be calculated for one participant. | 0.65 (NA) — Standard deviation could not be calculated for one participant. | 0.50 (NA) — Standard deviation could not be calculated for one participant. | 1.13 (NA) — Standard deviation could not be calculated for one participant.
  Day 14: 20 minutes- Corner,n=1,1,1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1
  Day 14: 20 minutes- Corner,n=1,1,1,1,1,1,1 | 0.50 (NA) — Standard deviation could not be calculated for one participant. | 1.87 (NA) — Standard deviation could not be calculated for one participant. | 8.54 (NA) — Standard deviation could not be calculated for one participant. | 0.36 (NA) — Standard deviation could not be calculated for one participant. | 0.30 (NA) — Standard deviation could not be calculated for one participant. | 0.50 (NA) — Standard deviation could not be calculated for one participant. | 0.50 (NA) — Standard deviation could not be calculated for one participant.
  Day 14: 20 minutes- Bench,n=1,1,1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1
  Day 14: 20 minutes- Bench,n=1,1,1,1,1,1,1 | 0.50 (NA) — Standard deviation could not be calculated for one participant. | 1.39 (NA) — Standard deviation could not be calculated for one participant. | 6.47 (NA) — Standard deviation could not be calculated for one participant. | 0.27 (NA) — Standard deviation could not be calculated for one participant. | 0.50 (NA) — Standard deviation could not be calculated for one participant. | 0.50 (NA) — Standard deviation could not be calculated for one participant. | 0.50 (NA) — Standard deviation could not be calculated for one participant.
  Day 1: 60 minutes- Corner,n=1,1,1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1
  Day 1: 60 minutes- Corner,n=1,1,1,1,1,1,1 | 0.89 (NA) — Standard deviation could not be calculated for one participant. | 0.13 (NA) — Standard deviation could not be calculated for one participant. | 0.99 (NA) — Standard deviation could not be calculated for one participant. | 2.03 (NA) — Standard deviation could not be calculated for one participant. | 2.34 (NA) — Standard deviation could not be calculated for one participant. | 0.10 (NA) — Standard deviation could not be calculated for one participant. | 0.10 (NA) — Standard deviation could not be calculated for one participant.
  Day 1: 60 minutes- Bench,n=1,1,1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1
  Day 1: 60 minutes- Bench,n=1,1,1,1,1,1,1 | 0.75 (NA) — Standard deviation could not be calculated for one participant. | 0.15 (NA) — Standard deviation could not be calculated for one participant. | 0.90 (NA) — Standard deviation could not be calculated for one participant. | 2.09 (NA) — Standard deviation could not be calculated for one participant. | 2.17 (NA) — Standard deviation could not be calculated for one participant. | 0.10 (NA) — Standard deviation could not be calculated for one participant. | 0.10 (NA) — Standard deviation could not be calculated for one participant.
  Day 7: 60 minutes- Corner,n=1,1,1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1
  Day 7: 60 minutes- Corner,n=1,1,1,1,1,1,1 | 0.22 (NA) — Standard deviation could not be calculated for one participant. | 1.72 (NA) — Standard deviation could not be calculated for one participant. | 1.19 (NA) — Standard deviation could not be calculated for one participant. | 0.19 (NA) — Standard deviation could not be calculated for one participant. | 0.34 (NA) — Standard deviation could not be calculated for one participant. | 0.10 (NA) — Standard deviation could not be calculated for one participant. | 0.46 (NA) — Standard deviation could not be calculated for one participant.
  Day 7: 60 minutes- Bench,n=1,1,1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1
  Day 7: 60 minutes- Bench,n=1,1,1,1,1,1,1 | 1.22 (NA) — Standard deviation could not be calculated for one participant. | 1.40 (NA) — Standard deviation could not be calculated for one participant. | 1.00 (NA) — Standard deviation could not be calculated for one participant. | 0.18 (NA) — Standard deviation could not be calculated for one participant. | 0.28 (NA) — Standard deviation could not be calculated for one participant. | 0.10 (NA) — Standard deviation could not be calculated for one participant. | 0.52 (NA) — Standard deviation could not be calculated for one participant.
  Day 14: 60 minutes- Corner,n=1,1,1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1
  Day 14: 60 minutes- Corner,n=1,1,1,1,1,1,1 | 0.10 (NA) — Standard deviation could not be calculated for one participant. | 0.70 (NA) — Standard deviation could not be calculated for one participant. | 3.58 (NA) — Standard deviation could not be calculated for one participant. | 0.10 (NA) — Standard deviation could not be calculated for one participant. | 0.14 (NA) — Standard deviation could not be calculated for one participant. | 0.10 (NA) — Standard deviation could not be calculated for one participant. | 0.10 (NA) — Standard deviation could not be calculated for one participant.
  Day 14: 60 minutes- Bench,n=1,1,1,1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1
  Day 14: 60 minutes- Bench,n=1,1,1,1,1,1,1 | 0.10 (NA) — Standard deviation could not be calculated for one participant. | 0.62 (NA) — Standard deviation could not be calculated for one participant. | 3.20 (NA) — Standard deviation could not be calculated for one participant. | 0.14 (NA) — Standard deviation could not be calculated for one participant. | 0.11 (NA) — Standard deviation could not be calculated for one participant. | 0.10 (NA) — Standard deviation could not be calculated for one participant. | 0.10 (NA) — Standard deviation could not be calculated for one participant.

73. Secondary Outcome: Part 1: Concentration of CCI15106 in Lung Epithelial Lining Fluid (ELF) in Repeated Dose of Cohort B 60 mg
Description: Bronchoalveolar lavage samples for ELF concentration analysis of CCI15106 were collected up to Day 13. Participants who received at least one dose of study treatment and who underwent bronchoalveolar lavage (BAL) sampling and had post-dose lung ELF CCI15106 and urea concentration result were included in BAL PK Population.
Time Frame: Up to Day 13
Population: BAL PK Population.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | Part 1: Cohort B- CCI15106 60 mg BID
Number analyzed (Participants) | 12
Nanogram per milliliter | 47306.383 (25231.0613)

74. Secondary Outcome: Part 2: Concentration of CCI15106 in ELF in Repeated Dose of Cohort B 60 mg
Description: BAL samples for ELF concentration analysis of CCI15106 were collected up to Day 13.
Time Frame: Up to Day 13
Population: BAL PK Population.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | Part 2: Cohort B- CCI15106 60 mg BID
Number analyzed (Participants) | 8
Nanogram per milliliter | 247290.327 (427471.7407)

75. Secondary Outcome: Part 1: Number of Participants With Medical Device Incidents in CCI15106
Description: A medical device incident is any malfunction or deterioration in the characteristics and/or performance of a device as well as any inadequacy in the labeling or the instructions for use which, directly or indirectly, might lead to or might have led to the death of a participant/user/other person or to a serious deterioration in his/her state of health.
Time Frame: Up to Day 19
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort A- CCI15106 60 mg SD | Part 1: Cohort A- CCI15106 120 mg SD | Part 1: Cohort A- CCI15106 30 mg BID | Part 1: Cohort B- CCI15106 60 mg BID | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 12 | 4
Participants | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected up to 51 days for Cohort A in Part 1, 46 days for Cohorts B and C in Part 1; 33 days for Cohort A in Part 2 and 46 days for Cohort B in Part 2
Description: Safety population was used to assess NSAEs and SAEs.
Arm/Group | Part 1: Cohort A- CCI15106 60 mg SD | Part 1: Cohort A- CCI15106 120 mg SD | Part 1: Cohort A- CCI15106 30 mg BID | Part 1: Cohort A- Placebo | Part 1: Cohort B- CCI15106 60 mg BID | Part 1: Cohort B- Placebo | Part 1: Cohort C- Bystanders | Part 2: Cohort A- CCI15106 60 mg SD | Part 2: Cohort A- Placebo | Part 2: Cohort B- CCI15106 60 mg BID
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/2 | 0/12 | 0/2 | 0/14 | 0/6 | 0/2 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/2 | 0/12 | 0/2 | 0/14 | 0/6 | 0/2 | 0/8
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/2 | 6/12 | 0/2 | 6/14 | 0/6 | 0/2 | 7/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Cohort A- CCI15106 60 mg SD (N=6) | Part 1: Cohort A- CCI15106 120 mg SD (N=6) | Part 1: Cohort A- CCI15106 30 mg BID (N=6) | Part 1: Cohort A- Placebo (N=2) | Part 1: Cohort B- CCI15106 60 mg BID (N=12) | Part 1: Cohort B- Placebo (N=2) | Part 1: Cohort C- Bystanders (N=14) | Part 2: Cohort A- CCI15106 60 mg SD (N=6) | Part 2: Cohort A- Placebo (N=2) | Part 2: Cohort B- CCI15106 60 mg BID (N=8)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-04-20): https://cdn.clinicaltrials.gov/large-docs/26/NCT03235726/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-30): https://cdn.clinicaltrials.gov/large-docs/26/NCT03235726/SAP_001.pdf